# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

DMID Protocol: 16-0073 Study Title:

A Randomized, Double-Blind, Placebo Controlled, Phase 2
Study to Assess Treatment of Gardnerella vaginalis
Vaginal Colonization with Amoxicillin
NCT03211156

Version 1.0

**DATE: 27-FEB-2019** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

#### STUDY TITLE

| <b>Protocol Number Code:</b> | DMID Protocol: 16-0073 |
|---|---|
| <b>Development Phase:</b> | Phase 2 |
| Products: | Amoxicillin |
| Form/Route: | Oral |
| Indication Studied: | Gardnerella vaginalis |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | 21SEP2017 |
| Clinical Trial Completion Date: | TBD |
| Date of the Analysis Plan: | 27FEB2019 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | II |
|---|---|---|
| TABLE | OF CONTENTS | III |
| LIST O | F ABBREVIATIONS | VI |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 2.1. | Purpose of the Analyses | 2 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. | Study Objectives | 3 |
| 3.2. | Endpoints | 3 |
| 3.3. | Study Definitions and Derived Variables | 3 |
| 3.3.1. | BV Diagnosis by Amsel Criteria | 3 |
| 3.3.2. | Nugent Criteria for Determination of BV | 3 |
| 3.3.3. | Eradication of GV | 4 |
| 3.3.4. | GV Positive | 4 |
| 3.3.5. | Evaluable | 4 |
| 3.3.6. | Treatment Compliance | 4 |
| 3.3.7. | Baseline value | 4 |
| 3.3.8. | Test of Cure Visit | 4 |
| 4. | INVESTIGATIONAL PLAN | 5 |
| 4.1. | Overall Study Design and Plan | 5 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 5 |
| 4.3. | Selection of Study Population | 6 |
| 4.4. | Treatments | 7 |
| 4.4.1. | Treatments Administered | 7 |
| 4.4.2. | Identity of Investigational Product(s) | 7 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 7 |
| 4.4.4. | Selection of Doses in the Study | 8 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 8 |
| 4.4.6. | Blinding | 8 |
| 4.4.7. | Prior and Concomitant Therapy | 8 |

# **Table of Contents** (continued)

| 4.4.8. | Treatment Compliance | 9 |
|----------|------------------------------------------------|----|
| 4.5. | Efficacy and Safety Variables | 9 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 11 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 12 |
| 6.1. | General Principles | 12 |
| 6.1.1. | Pseudo Code | 12 |
| 6.2. | Timing of Analyses | 13 |
| 6.3. | Analysis Populations | 13 |
| 6.3.1. | Safety Analyses | 13 |
| 6.3.2. | Efficacy Analyses | 13 |
| 6.3.2.1. | Intent-to-Treat (ITT) Population | 13 |
| 6.3.2.2. | NAAT Screening Population | 13 |
| 6.3.2.3. | Per-Protocol Population | 13 |
| 6.3.3. | Analysis Population Summaries | 14 |
| 6.4. | Covariates and Subgroups | 14 |
| 6.5. | Missing Data | 14 |
| 6.6. | Interim Analyses and Data Monitoring | 14 |
| 6.7. | Multicenter Studies | 15 |
| 6.8. | Multiple Comparisons/Multiplicity | 15 |
| 7. | STUDY SUBJECTS | 16 |
| 7.1. | Disposition of Subjects | 16 |
| 7.2. | Protocol Deviations | 16 |
| 8. | EFFICACY EVALUATION | 17 |
| 8.1. | Primary Efficacy Analysis | 17 |
| 8.2. | Secondary Efficacy Analyses | 17 |
| 8.3. | Exploratory Efficacy Analyses | 17 |
| 9. | SAFETY EVALUATION | 19 |
| 9.1. | Demographic and Other Baseline Characteristics | 19 |
| 9.1.1. | Prior and Concurrent Medical Conditions | 19 |
| 9.1.2. | Prior and Concomitant Medications | 19 |
| 9.2. | Measurements of Treatment Compliance | 19 |

# **Table of Contents** (continued)

| 9.3. | Adverse Events | 20 |
|---|---|---|
| 9.3.1. | Solicited Events and Symptoms | 20 |
| 9.3.2. | Unsolicited Adverse Events | 20 |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 21 |
| 9.5. | Pregnancies | 21 |
| 9.6. | Clinical Laboratory Evaluations | 21 |
| 9.7. | Vital Signs and Physical Evaluations | 21 |
| 10. | PHARMACOKINETICS | 22 |
| 11. | IMMUNOGENICITY | 23 |
| 12. | OTHER ANALYSES | 24 |
| 13. | REPORTING CONVENTIONS | 25 |
| 14. | TECHNICAL DETAILS | 26 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 27 |
| 16. | REFERENCES | 28 |
| 17. | LISTING OF TABLES, FIGURES, AND LISTINGS | 29 |
| APPENI | DICES | 30 |
| APPENI | DIX 1. TABLE MOCK-UPS | 31 |
| APPENI | DIX 2. FIGURE MOCK-UPS | 83 |
| APPENI | DIX 3. LISTINGS MOCK-UPS | 88 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|--------------------------------------------------|
| BV | Bacterial Vaginosis |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data Safety Monitoring Board |
| EDC | Electronic Data Capture |
| FDA | Food and Drug Administration |
| GV | Gardnerella vaginalis |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonisation |
| IDES | Internet Data Entry System |
| ISM | Independent Safety Monitor |
| ITT | Intention to Treat |
| КОН | Potassium hydroxide |
| LLOQ | Lower Limit of Quantification |
| ULOQ | Up Limit of Quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| N | Number (typically refers to subjects) |
| NAAT | Nucleic Acid Amplification Test |
| NIH | National Institutes of Health |
| pН | Potential of Hydrogen |
| PI | Principal Investigator |
| PO | Per os (by mouth) |
| PP | Per Protocol |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |

# **List of Abbreviations** (continued)

| SD | Standard Deviation |
|------|------------------------------------------|
| SDCC | Statistical and Data Coordinating Center |
| SOC | System Organ Class |
| STD | Sexually transmitted disease |
| TOC | Test of Cure |
| UAB | University of Alabama at Birmingham |
| USP | United States Pharmacopeia |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Randomized, Double-Blind, Placebo Controlled, Phase 2 Study to Assess Treatment of Gardnerella vaginalis Vaginal Colonization with Amoxicillin" (DMID Protocol 16-0073) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA) and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for efficacy and safety outcomes, and (4) a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Bacterial Vaginosis (BV) is the most common cause of vaginitis worldwide and is strongly associated with important public health issues including preterm birth and acquisition/transmission of Human Immunodeficiency Virus (HIV) and other sexually transmitted diseases (STDs) [reference 1-2 in protocol]. Although the exact cause of BV is unclear, the current epidemiologic data strongly support the hypothesis that BV is sexually transmitted [reference 3 in protocol]. Further, there is mounting data to suggest that Gardnerella vaginalis (GV) is the founder organism that is sexually transmitted [reference 3 in protocol]. Once GV is established, there is a resultant change in the vaginal microbiome characterized by loss of lactobacilli and an increase in anaerobic organisms leading to the syndrome of BV [reference 3-4 in protocol]. GV is nearly universally found in women with BV. However, it may also be found in women who do not meet the current definition of BV, leading some to question its pathogenicity. Others have hypothesized that there are strain differences among GV in terms of virulence factors [reference 5 in protocol].

If GV is necessary for the development of BV, then eradication of GV in women who do not meet the clinical criteria for BV should abort the future development of BV. Amoxicillin was chosen as the therapeutic intervention because it is highly active against GV but has limited efficacy against anaerobes associated with BV. This Phase 2 study will determine if GV in the vaginal flora will be eradicated by amoxicillin. If amoxicillin successfully eradicates GV, we will develop the next step to examine prevention of BV through screening and treatment of GV.

#### 2.1. Purpose of the Analyses

These analyses will assess the efficacy and safety of Amoxicillin in comparison with the placebo and will be included in the CSR.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

Primary Objective:

• To determine if treatment with amoxicillin eradicates GV in women who are colonized/infected with GV but have no clinical evidence of BV.

Secondary Objective:

• To evaluate the safety and tolerability of amoxicillin compared to placebo.

**Exploratory Objectives:** 

• To determine the demographic and behavioral factors associated with vaginal colonization of GV.

# 3.2. Endpoints

Primary Endpoint:

• The proportion of participants with eradication of GV in each study arm at Visit 2 (Day 15-21) as assessed by nucleic acid amplification test (NAAT).

Secondary Endpoint:

• The proportion of participants reporting related adverse events (AEs) and serious adverse events (SAEs) in each study arm following the first dose of study product through Visit 2 (Day 15-21).

**Exploratory Endpoint:** 

• The demographic and behavioral factors among women in the NAAT screening population without vaginitis who are baseline GV positive and women who are baseline GV negative.

# 3.3. Study Definitions and Derived Variables

#### 3.3.1. BV Diagnosis by Amsel Criteria

During pelvic examination, a positive clinical diagnosis of BV by Amsel criteria is defined as the presence of:

- 1) A fishy odor of the vaginal discharge with the addition of a drop of 10% potassium hydroxide (KOH) (positive whiff test); and
- 2) Clue cells  $\geq 20\%$  of the total vaginal squamous epithelial cells on saline microscopy; and
- 3) Vaginal fluid pH > 4.5.

If a subject does not meet at least one of the above criteria, then the clinical diagnosis of BV is negative.

#### 3.3.2. Nugent Criteria for Determination of BV

The Nugent score utilizes a 0-10 point scale for evaluation of vaginal flora and is based on the weighted sum score of the following three bacterial morphotypes calculated from the slide exam under oil immersion (1000x):

- Lactobacillus: Large Gram-negative rods
- Gardnerella/Bacteroides spp: thin, curved, Gram-variable rods

#### • Mobiluncus spp: thin, curved, Gram-variable rods

The Nugent score is interpreted as follows: 0-3 normal; 4-6 intermediate; and 7-10 BV. For the purposes of this study, a score > 3 is considered abnormal, and a score of 0-3 is considered normal.

#### 3.3.3. Eradication of GV

Eradication of GV is defined by a negative NAAT result for GV at Visit 2 (Day 15-21).

#### 3.3.4. GV Positive

Any subjects with NAAT results of valid numeric values including "< LLOQ" and ">ULOQ" are considered positive for GV.

#### 3.3.5. Evaluable

Participants are deemed evaluable if their BV and GV status can be determined at screening and their GV status can be determined at Visit 2. Participants who are missing Gram stain, GV NAAT, or Amsel results at screening are not evaluable. Participants who are missing GV NAAT results at the Visit 2 are not evaluable.

#### 3.3.6. Treatment Compliance

A participant is considered adherent to the study treatment regimen if she uses at least 80% of the scheduled doses (i.e. at least 12 of the 14 doses) of study treatment, as assessed by the number of pills returned. If pill count cannot be assessed, participant report will be used to assess adherence.

#### 3.3.7. Baseline value

The baseline value will be defined as the last value obtained prior to the first dose of study product.

#### 3.3.8. Test of Cure Visit

The test of cure (TOC) visit is defined as the Visit 2 (Day 15-21) visit.

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

This is a randomized, double-blind, placebo-controlled Phase 2 study screening approximately 245 adult females 18-45 years of age to enroll approximately 98 participants to achieve 82 evaluable participants at the test of cure (TOC) visit. The study is designed to determine if amoxicillin will eradicate vaginal colonization/infection with GV when administered to women who are colonized/infected with GV but have no clinical evidence of BV. Women who consent to screening participation undergo pelvic examination on entry and vaginal specimens collected for pH, whiff test and wet prep microscopy (Amsel criteria with the exception of evaluation of vaginal discharge), Nugent score, NAAT for trichomonas, and quantitative NAAT for GV. At Visit 1 (Enrollment - Day 1) women who tested positive for GV by NAAT, negative for BV by Nugent and negative for trichomonas by NAAT are enrolled and randomized to one of two groups (amoxicillin or placebo). A TOC is completed at Visit 2 (Day 15-21).

Baseline information is collected from all women at the screening visit (Visit 0 (Day -14 to -7). This information consists of demographics, medical and sexual history, concomitant medications, and clinical and laboratory findings. Vaginal swabs are collected as noted above. Women who test positive for vaginitis at the screening visit are screen failures. At the Enrollment Visit (Visit 1, Day 1) women who tested positive for GV, negative for abnormal flora/BV, and negative for trichomonas are enrolled and randomized. Those who were negative for GV are screen failures and do not continue in the study, but, their, demographic, medical, and sexual history as well as baseline swabs are used for comparisons to the GV positive women for an exploratory objective.

Women who are enrolled are asked to return for one further visit, Visit 2 (Day 15-21), where a TOC is completed (a pelvic exam completed with the same specimens taken as those at baseline with the exception of the trichomonas NAAT).

Participants are queried regarding any adverse outcomes and all AEs will be collected through Visit 2. Laboratory testing includes (NAAT for trichomonas; Nugent score for BV; quantitative NAAT for GV; and assessment of vaginal pH, saline microscopy (yeast, trichomonas, clue cells).

The duration of the study for participants who are enrolled and randomized is approximately 22 days. For those not enrolled, participation ends at their post screening follow up phone call.

Safety oversight is provided by an Independent Safety Monitor (ISM) at each clinical site and by a Data Monitoring Safety Board (DSMB). The DSMB members meets at specified times during the course of the study as defined in the DSMB Charter.

Table 1 presents the schematic of the study design and Table 2 presents the schedule of study procedures.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

This phase 2 study is designed to determine if amoxicillin will eradicate GV in the vaginal flora. The assumption is that GV is necessary for the development of BV, so eradication of GV in women who do not meet the clinical criteria for BV should halt future development of BV. Amoxicillin was chosen due to its highly active therapeutic response to GV, but also due to its limited efficacy against anaerobes associated with BV. If this study shows that amoxicillin successfully eradicates GV, then the next step will be to examine whether screening and treatment of GV will prevent BV. Participants are randomized using a 1:1 ratio to receive amoxicillin or placebo.

# 4.3. Selection of Study Population

Women eligible to enroll in this this study must meet all of the inclusion criteria:

- 1. Women ages 18-45, inclusive;
- 2. No evidence of vaginitis (yeast, trichomonas, and BV/abnormal vaginal flora) or other vaginal conditions which in the opinion of the investigator could be confounders\*;
  - \*These causes will initially be detected by wet mount microscopy with trichomonas during the screening procedures and later confirmed by NAAT and BV/abnormal vaginal flora confirmed by Nugent scoring (Nugent score of 4-10);
- 3. Presence of GV detected by NAAT\*;
  - \*results of NAAT testing will be available prior to return for Enrollment visit;
- 4. Willing to use condoms during vaginal intercourse while participating in the study;
- 5. Not currently menstruating at screening visit;
- 6. Willing and able to provide written informed consent;
- 7. Negative urine pregnancy test on all participants of childbearing potential at study screening;
- 8. Participant must be of non-childbearing potential\* or must be using highly effective birth control\*\* to avoid becoming pregnant.
  - \*Non-childbearing potential is defined as being post-menopausal for at least 1 year, status after bilateral tubal ligation, or status after bilateral oophorectomy or status after hysterectomy.
  - \*\*In addition to the required use of condoms by the male partner during study participation, participants must agree to avoid becoming pregnant by using one of the following acceptable methods of birth control for 30 days prior to screening and for the duration of the study;
    - Intrauterine contraceptive device; OR
    - Oral contraceptives; OR
    - Hormonal injections; OR
    - Hormonal implants; OR
    - Contraceptive patches; OR
    - Monogamous relationship with vasectomized partner; OR
    - Exclusively same-sex relationships; OR
    - Abstinence:
- 9. Participant is not planning on taking antibiotics or using any intravaginal microbicides from the Screening visit through the Visit 2 Follow-up (TOC);
- 10. Participant is willing and able to cooperate to the extent and degree required by this protocol at the discretion of the investigator.

Participants eligible to participate in this study must not meet any of the following exclusion criteria:

1. Pregnant or nursing:

- 2. Allergic to penicillin, amoxicillin, cephalosporins, or other β-lactam antibiotic;
- 3. Use of antibiotics in the past 14 days prior to screening visit;
- 4. HIV infected;
- 5. Women taking immunosuppressive agents;
- 6. History of renal impairment;
- 7. Use of any investigational drug within the past 30 days prior to screening;
- 8. Any other condition that, in the opinion of the investigator, would interfere with participation in the study.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Participants are randomized using a 1:1 ratio to receive amoxicillin or placebo.

The dates of first treatment are presented for subjects in the Safety population by site in Table 3 and actual treatment group in Table 4.

#### 4.4.2. Identity of Investigational Product(s)

#### **Amoxicillin**

Amoxicillin, United States Pharmacopeia (USP) is a semisynthetic antibiotic, an analog of ampicillin, with a broad spectrum of bactericidal activity against many gram-positive and gram-negative microorganisms. Amoxicillin is similar to penicillin in its bactericidal action against susceptible bacteria during the stage of active multiplication. It acts through the inhibition of cell wall biosynthesis that leads to the death of the bacteria.

Amoxicillin will be supplied as 250 mg amoxicillin trihydrate. Each active capsule of amoxicillin will be placed in a gelatin capsule. The gelatin capsules are Swedish orange capsules from Capsugel. Each vial contains 28 capsules.

#### Placebo for Amoxicillin

Each placebo capsule will be filled with lactose only and will be identical in appearance to the capsule with the active ingredient. The lactose filler is Lactose USP and the small amount should not be a problem even for persons who are lactose-intolerant. Participants may experience some mild bloating. Each vial contains 28 capsules

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment of participants is done online using the enrollment module of AdvantageEDC<sup>SM</sup>. Participants are randomized using a 1:1 ratio to receive amoxicillin or placebo after providing consent and confirmation of eligibility based on the study inclusion and exclusion criteria. The study uses a stratified, permuted block randomization scheme. Permuted block randomization is used to avoid the potential for serious imbalance in the number of participants assigned to each group, an imbalance that can occur in the simple randomization procedures. Stratification is by study site.

The list of randomized treatment assignments is prepared by statisticians at the Emmes Corporation and provided to the research pharmacist at University of Alabama at Birmingham (UAB) who will prepare the study treatment. The research pharmacist will label each vial of study treatment with a blinded treatment number according to the randomization scheme. The list of randomized treatment assignments is included in the enrollment module of The Emmes Corporation's Internet Data Entry System (IDES). IDES assigns each enrolled participant a blinded vial number after demographic and eligibility data have been entered into the system.

Each site has a supply of blinded vials pre-labeled with treatment numbers, each containing sufficient doses to treat a participant for seven days. Once a participant is assigned a vial number, the vial is distributed to the participant.

#### 4.4.4. Selection of Doses in the Study

Participants are randomized to one of two study products as follows:

- Amoxicillin 2 x 250mg capsules PO twice a day for 7 days
- Placebo 2 capsules PO twice a day for 7 days

#### 4.4.5. Selection and Timing of Dose for Each Subject

At the enrollment visit, Visit 1, subjects that are eligible to receive treatment will be randomized (1:1 ratio) to receive either amoxicillin or placebo. Each subject will receive 14 doses (2 x 250mg capsules) of amoxicillin or placebo to be taken orally, twice a day, for 7 consecutive days. The first dose should be taken in the evening after the enrollment visit. The subject should then take one dose in the morning and one dose in the evening for the next seven days. Subjects should take the doses approximately 12 hours apart. Only one dose is taken on the morning of the eighth day.

#### 4.4.6. Blinding

Amoxicillin and placebo are masked by providing identical study vials to participants in the two arms. All participants and clinical investigators participating in this trial are blinded with respect to treatment assignment. The research pharmacy at UAB over-encapsulates the amoxicillin capsules for the active treatment arm and creates identical appearing placebo capsules containing lactose.

The participants, the study personnel who perform study assessments after administration and those dispensing study medication, data entry personnel at the sites, and laboratory personnel are blinded to treatment assignment. The DSMB may receive data in aggregate and presented by treatment group, but without the treatment group identified. The DSMB may be unblinded to individual study treatment assignments, as needed, to adequately assess safety issues.

The protocol contains no explicit provisions for emergency unblinding. According to DMID policy, the study medical monitor responds to requests for emergency unblinding and instructs the Statistical and Data Coordinating Center (SDCC) to release treatment codes only if necessary to ensure that the subject receives appropriate clinical care.

#### 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines are recorded on the appropriate data collection form. Concomitant medications include all medications taken 14 days prior to the screening visit through Visit 2 or early termination, whichever occurs first. Prescription and over-the-counter drugs are included, as

well as intravaginal products, herbs, vitamins, and supplements. Previously recorded medications are updated as appropriate. Assessment of eligibility also includes a review of all permitted and prohibited medications per the participant inclusion and exclusion criteria (See Section 4.3).

Participants who have received study drug and are subsequently diagnosed with a concomitant infection that requires systemic antibiotics receive treatment according to the local clinic's standard protocols.

Medications that might interfere with the evaluation of the treatment should not be used unless absolutely necessary. Medications in this category include, but are not limited to, antibiotics and intravaginal microbicides.

#### 4.4.8. Treatment Compliance

Participants are instructed to record the date and timing of all doses on a memory aid. Participants are asked to bring the vial of medication and memory aid to the study personnel at their follow-up visit. Study personnel reviews adherence to the study medication schedule with the participants, including the participant's memory aid, and record this on the appropriate data collection form at Visit 2 (TOC). See Section 3.3.5 for the definition of adherence to treatment.

#### 4.5. Efficacy and Safety Variables

For safety and efficacy analyses, multiple observations within a specific visit period are accepted. In the case of multiple observations within a specific window, the assessment value that is closest to the scheduled visit window will be used in the analyses for the post-baseline records. For screening and baseline visits, the last assessment value will be used. All the recorded data will be listed. If observations have the same distance to the scheduled assessment, the latest one will be used.

#### **Efficacy Variables**

See Section 3.3 for efficacy variable definitions. Eradication of GV is the primary efficacy variable. Amsel criteria and Nugent scores will be determined to diagnose BV according to the definition in Section 3.3. See Section 3.3 for efficacy variable definitions. BV recurrence is the primary efficacy variable. Amsel criteria and Nugent scores will be determined at each follow-up visit to diagnose BV according to the definition in Section 3.3.1.

#### **Safety Variables**

#### Adverse Event

ICH E6 defines an AE as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal product. AEs will be graded using the following general criteria:

- Mild: events require minimal or no treatment and do not interfere with the patient's daily activities.
- Moderate: events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
- Severe: events interrupt a patient's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually incapacitating.

#### Serious Adverse Event

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death,
- a life-threatening adverse event,
- inpatient hospitalization or prolongation of existing hospitalization,
- a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
- a congenital anomaly/birth defect.
- Important medical events that may not result in death, be life-threatening, or require hospitalizations may be considered serious when, based upon appropriate medical judgment they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 5. SAMPLE SIZE CONSIDERATIONS

Sample size calculations were based on detecting a decrease in GV colonization rate from 80% among participants receiving placebo to as large as 44% among participants receiving amoxicillin. Using the two-sided Pearson Chi-Square test with Yates continuity correction, significance level of 0.05, and assuming an amoxicillin to placebo allocation ratio of 1:1, 82 women (41 in each arm) would provide 90% power to detect a difference in colonization rates of 36% (i.e. 44% colonization rate in the amoxicillin arm).

Assuming a 15% drop-out rate between enrollment and the TOC visit approximately 98 women will need to be randomized to obtain 82 women evaluable for the primary analysis. Assuming 40% of women without BV will have a positive NAAT test for GV at screening, approximately 245 women without BV will need to be screened to randomize 98 women in the study.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

#### **6.1.** General Principles

Tabulations will be used extensively to summarize the data. All continuous variables will be summarized using the following descriptive statistics: n (sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the sample size) of observed levels will be reported for all categorical measures. Wilson confidence intervals for binomial proportions and differences in binomial proportions will be computed for efficacy variables. Blaker confidence intervals for binomial proportions and differences in binomial proportions will be computed for safety variables. For the hypothesis tests comparing treatment groups with respect to safety outcomes, the two-sided Fisher's Exact test will be used. For the hypothesis tests comparing treatment groups with respect to efficacy outcomes, the two-sided Pearson Chi-Square test with Yates continuity correction will be used. For all tests, a 5% two-sided significance level will be used.

For all efficacy outcome measures, the Intention-to-Treat (ITT) population (see Section 6.3) will be used as the primary analysis population and the Per Protocol population will be used as a secondary analysis population. For all safety analyses, the Safety population will be used as the analysis population.

All summary tables will be structured with a column/sub-table for each treatment group (Amoxicillin, Placebo, and All Subjects). In general, all data will be listed by treatment group and/or subject, and when appropriate by visit number within subject. The total population size relevant to that table/column if applicable, including any missing observations will be displayed in the tables.

Note that in the data listings, Subject ID is the unique subject identifier, not the Study ID used on study and dates will not be included, only Study Day.

#### 6.1.1. Pseudo Code

The following SAS® pseudo code will be used to calculate the following:

Chi-Square test at 5% two-sided significance level and odds ratio (and 95% asymptotic CI) from 2x2 table:

```
proc freq;
      Table treatment*analysis variable / chisq;
      ods output ChiSq=outputdsn1;
      ods output RelativeRisks=outputdsn2;
run;
Note: Yates continuity correction is where Statistic = "Continuity Adj. Chi-Square";
Fisher's Exact test at 5% two-sided significance level:
proc freq;
      Table treatment*analysis variable / exact;
      ods output FishersExact=outputdsn;
run:
95% Wilson CI for proportions/percentages:
proc freq;
      Table treatment*analysisvariable / binomial(wilson);
      ods output binomialcls=outputdsn;
run;
```

95% Wilson CI for difference in proportions (produces Newcombe CI):

```
proc freq;
        Table treatment*analysisvariable / riskdiff(cl=Wilson);
        Exact Riskdiff;
        ods output pdiffcls=outputdsn;
run;

95% Exact Blaker CI for proportions/percentages:
proc freq;
        Table treatment*analysisvariable / binomial(blaker);
        ods output binomialcls=outputdsn;
run;
```

#### **6.2.** Timing of Analyses

The final analysis will be performed after database lock when all subjects have been followed through Visit 2, the final study visit, at Day 15 (Window: Days 15-21).

#### 6.3. Analysis Populations

#### **6.3.1.** Safety Analyses

All safety analyses will be performed in the Safety population. The Safety population includes all randomized subjects who received at least one dose of treatment. In the unlikely event of an error in randomization or treatment administration (i.e., incorrect product), subjects will be grouped by the product they actually received.

#### **6.3.2.** Efficacy Analyses

All efficacy analyses will be performed in the Intent-to-Treat (ITT) and Per Protocol (PP) analysis populations. The NAAT screening population will be used as the exploratory efficacy analysis population.

#### 6.3.2.1. Intent-to-Treat (ITT) Population

The ITT population includes all randomized subjects, regardless of whether they received study treatment or were compliant with the administration procedures or schedule. In the unlikely event of an error in randomization or treatment administration (i.e., incorrect product), subjects will be grouped by their intended randomized assignment.

#### **6.3.2.2.** NAAT Screening Population

The NAAT Screening population includes all screened women who are evaluated for GV by NAAT.

#### 6.3.2.3. Per-Protocol Population

The PP population includes all randomized participants who met all inclusion/exclusion criteria, are evaluable, adhered to the assigned study treatment regimen (as defined in Section 3.3.5), and returned to the study site for the TOC visit within the specified window (Visit 2 [Window: Day 15 -21]) and did not experience any of the following after enrollment:

• Unprotected vaginal sexual intercourse between Visit 1 and Visit 2

- New pregnancy reported by the subject
- Receipt of any antibiotic or intravaginal microbicide other than study drug

In the unlikely event of an error in randomization or treatment administration (i.e., incorrect product), subjects will be grouped by the product they actually received.

#### **6.3.3.** Analysis Population Summaries

Table 5 summarizes the Safety and PP population eligibilities by actual treatment group and reasons excluded. Subjects will be included in the count for a particular reason for Exclusion if they met that criterion. As subjects may meet more than one criterion for exclusion, the "Excluded from..." counts may be less than the sum of the individual reason counts. A listing of the subjects excluded from each of the analysis populations and the reasons for exclusion will be provided (Listing 1). A listing of subjects whose assigned treatment group does not match their randomized treatment group will be provided in Listing 2.

#### 6.4. Covariates and Subgroups

The protocol does not define any subgroup analyses for the primary and secondary efficacy analyses, while the exploratory efficacy analysis will be performed within subgroups defined by demographic and baseline characteristics of participants. Safety and enrollment summaries will be presented by clinical site.

# 6.5. Missing Data

Subjects who are not evaluable will be excluded from the PP population.

Participants who have a missing GV NAAT result at the TOC visit are excluded from the PP analyses. For the ITT population, participants who have a missing GV NAAT result at the TOC visit will be classified as treatment failures.

For ITT population, the Worst-Case imputation will also be explored. In this analysis, participants who have a missing GV NAAT result at the TOC visit in Amoxicillin arm will be classified as treatment failures while those who in placebo arm will be classified as cures.

Only GV eradication status will be imputed.

# 6.6. Interim Analyses and Data Monitoring

The study is monitored to determine if the following safety halting rule is met:

1) If any two participants experience an adverse event that is judged to be Severe (Grade 3) and related to treatment

If the halting rule is met, the study will not continue with the remaining enrollments or study treatments without a review by and recommendation from the DSMB to proceed. A summary of subjects meeting the halting rule is provided in Table 6. The DSMB may review study progress and participant safety data at study specific time frames, at least annually, as defined in the DSMB Charter. The halting rule does not utilize any statistical criteria and no formal hypothesis testing is planned to occur for the safety and enrollment data reviews.

# 6.7. Multicenter Studies

Safety and efficacy data will be pooled across all clinical sites. Center effects are not anticipated because treatment is self-administered, the sites are using standardized procedures for assessment of unsolicited adverse events, and the study relies on a central laboratory for Quantitative NAATs and Gram stain Nugent scoring.

# 6.8. Multiple Comparisons/Multiplicity

No adjustments for multiple testing are planned.

#### 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

Table 7 shows the number of subjects who are screen failures, the number of subjects that met each inclusion/exclusion criterion, and the number of subjects who were eligible but declined enrollment. The number of enrolled subjects in the study completing study milestones will be tabulated separately by randomized treatment group and all subjects. Table 8 shows the total number of subjects screened, enrolled or randomized, treated, complying with treatment, and completing the TOC visit (Visit 2). A listing of subjects who completed the study, terminated early from study, or discontinued treatment and the reason for early termination or treatment discontinuation is included in Listing 3.

Figure 1 is a flowchart showing the disposition of study subjects in the safety and efficacy analyses, adapted from the CONSORT statement [1]. It shows the number of subjects eligible, enrolled and randomized, lost to follow-up, and analyzed for the safety, ITT and PP analyses by treatment group.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the deviation category, the type of deviation, and randomized treatment group for all enrolled subjects (Table 9). All subject-specific protocol deviations and non-subject-specific protocol deviations will be included in Appendix 3 as data listings (Listing 4 and Listing 5, respectively).

#### 8. EFFICACY EVALUATION

# 8.1. Primary Efficacy Analysis

The primary efficacy endpoint is the proportion of subjects with eradication of GV in each study arm at Visit 2 (Day 15-21) as assessed by NAAT. See Section 3.3.3 for the definition of eradication.

A test of hypothesis comparing the proportion of subjects with eradication of GV at Visit 2 (Day 15-21), will be conducted in the ITT population using the randomized treatment, and repeated as a secondary analysis using the actual treatment received in the PP population. The null hypothesis for each comparison is that there is no difference in proportions between treatment groups, with a two-sided alternative that considers the possibility of a difference in either direction. The test will be conducted using a Pearson Chi-Square test with Yates continuity correction at the 5% two-sided significance level. The number of subjects, the proportion of subjects with eradication of GV, and the 95% Wilson confidence interval for the proportion of subjects with eradication of GV will be presented for each analysis population and treatment group. In addition, the difference in proportions between the amoxicillin group and the placebo group and 95% Wilson confidence intervals will be presented. See Table 10 and Table 11. See Section 6.1 for pseudocode to fit the above analyses. Individual efficacy response data is presented in Listing 6.

# 8.2. Secondary Efficacy Analyses

There are no secondary efficacy objectives in this study.

#### **8.3.** Exploratory Efficacy Analyses

A summary of Amsel criteria is provided for subjects by visit and treatment group for each analysis population in Table 12 and Table 13. The number of Amsel criteria present (0,1,2,3), pH (> 4.5, ≤4.5), Clue cells (≥20%, < 20%), and Amine ("whiff") test on KOH wet mount (Positive, Negative) will be summarized. A summary of Amsel criteria is provided for subjects by treatment group and GV eradication status at Visit 2 for subjects in the ITT population and PP population (Table 14 and Table 15). GV eradication status is categorized as "GV Eradicated." "GV Not Eradicated," "Not Evaluable." See Section 3.3 for the definition of evaluable. A subject listing of individual Amsel criteria will be provided in Listing 6.

Table 16 and Table 17 presents the proportion of subjects with Nugent score of 3 or less (normal), 4-6 (intermediate), and 7-10 (BV) in each treatment group at Screening and at Visit 2 (Day 15-21). Continuous Nugent scores will also be presented by analysis population, study visit, and treatment group in Table 18 and Table 19. A subject listing of Nugent scores will be presented in Listing 6. Raw Nugent scores are displayed graphically by visit, treatment group, and analysis population in Figure 2 and Figure 3. Categorical and Continuous Nugent Score characteristics at Visit 2 are presented by GV eradication status, and treatment group for subjects in the ITT population and PP population (Table 20, Table 21, Table 22 and Table 23).

The mean count of *Lactobacillus spp.*, *Gardnerella/Bacteroides spp.*, and *Mobiluncus spp.*, respectively, in each treatment group at Screening and at Visit 2 (Day 15-21). Mean count and standard deviation of each specimen type will be presented by study visit, analysis population, and treatment group. Additionally, mean change from baseline and corresponding standard deviation will be presented for Visit 2. See Table 24 and Table 25. Mean count and standard deviation of *Lactobacillus spp.*, *Gardnerella/Bacteroides spp.*, and *Mobiluncus spp.* at Visit 2 is presented by GV eradication status for subjects in the ITT population and PP population (Table 26 and Table 27).

The exploratory outcome measure is the demographic and behavioral factors among women in the NAAT screening population without vaginitis who are baseline GV positive and women who are baseline GV negative. Gender, ethnicity, and race will be summarized by baseline GV status for subjects in the NAAT screening population in Table 28. Age will be summarized by baseline GV status in Table 29. Baseline GV status will be "Positive" or "Negative" as determined by NAAT at the screening visit.

Categorical and continuous sexual history questions will be summarized by baseline GV status (Table 30, Table 31) and by treatment group at baseline and Visit 2 BV status, respectively (Table 32, Table 33, Table 34, and Table 35)

Additionally, the demographic and baseline characteristics of participants who were positive for BV by Nugent Score and Amsel Criteria and by treatment group at Visit 2 (Day 15-21) will be summarized. See Table 36, Table 37, Table 38 and Table 39.

#### 9. SAFETY EVALUATION

# 9.1. Demographic and Other Baseline Characteristics

Demographic and other baseline characteristics will be summarized for all randomized subjects (ITT population). Gender, ethnicity, and race will be summarized by site (Table 40) and by randomized treatment group (Table 41). Ethnicity is categorized as Hispanic or Latino, or Not Hispanic or Latino. Race is categorized as American Indian or Alaska Native, Asian, Native Hawaiian or Other Pacific Islander, Black or African American, White, Multi-Racial, or Unknown. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race (Multi-Racial) or may refuse to identify a race (Unknown), the latter reflected in the Case Report Form (CRF) as "No" to each racial option. Age will be summarized by site (Table 42) and by randomized treatment (Table 43).

Baseline sexual history will be summarized for all randomized subjects (ITT population). Categorical sexual history questions will be summarized by treatment group (Table 44) and continuous sexual history questions will be summarized by treatment group (Table 45).

Individual subject listings will be presented for all demographics as well as baseline and follow-up sexual history for all enrolled subjects and GV negative Subjects respectively (Listing 8, Listing 9, Listing 10, Listing 11, Listing 12, Listing 13, Listing 14, Listing 15, Listing 16).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 20.1 or higher. Summaries of subjects' pre-existing and concurrent medical conditions will be presented by randomized treatment group for all sites and by each site in the ITT population (Table 46, Table 47, and Table 48).

Individual subject listings will be presented for all medical conditions (Listing 17).

#### 9.1.2. Prior and Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. Summaries of medications that were started prior to dosing and continuing at the time of dosing as well as medications that were started during dosing or during follow up will be presented by WHO Drug Anatomical Codes (ATC) Level 1 and Level 2 and actual treatment group for subjects in the Safety population (See Table 49, Table 50, and Table 51).

Individual subject listings will be presented for all concomitant medications and birth control methods (Listing 18 and Listing 19).

# **9.2.** Measurements of Treatment Compliance

All subjects are to receive a total of 14 doses of treatment. Each dose is to be taken orally, twice a day, for 7 consecutive days. Subjects should take the doses approximately 12 hours apart. See Section 3.3 and Section 4.4.8 for the definition of compliance that will be used for analyses.

The number of subjects not compliant with study treatment will be presented by treatment group as part of the subject disposition table (Table 8).

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the number of subjects in the safety population within the actual treatment group. All adverse events reported will be included in the summaries and analyses. All analyses in Section 9.3 will be performed in the safety analysis population using the actual treatment received.

#### 9.3.1. Solicited Events and Symptoms

Not applicable for this study.

#### 9.3.2. Unsolicited Adverse Events

The secondary endpoint is the proportion of subjects reporting related AEs and SAEs in each study arm following the first dose of treatment through Visit 2 (Day 15-21). The number of subjects, the proportion of subjects who experienced related AEs and SAEs following the first dose of treatment through Visit 2 (Day 15-21) and the 95% Blaker CIs for the proportion of subjects who experienced unsolicited AEs and SAEs related to treatment through Visit 2 will be presented for the safety population and actual treatment group. In addition, the difference in proportions between the Amoxicillin arm and the placebo arm and 95% Blaker CIs will be presented in Table 52.

The proportion of subjects who discontinue treatment early due to adverse events will be summarized overall and by treatment group. The number of subjects, the proportion of subjects who discontinue treatment early due to adverse events and the 95% Blaker CIs for the proportion will be presented for the safety population and actual treatment group. In addition, the difference in proportions between the Amoxicillin arm and the placebo arm and 95% Blaker CIs will be presented in Table 53.

The number of events and proportion of subjects reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term for all subjects and each actual treatment group. Denominators for percentages are the number of subjects who received the treatment being summarized. A 95% Blaker CI will be presented for each MedDRA system organ class and preferred term (Table 54). A subject listing of all adverse events is provided in Listing 20.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, and treatment group:

- The number and percentage of subjects by maximum severity and maximum relationship to treatment of events for all subjects and by actual treatment received (Table 55 and Table 56);
- The number of adverse events occurring in 5% of subjects in any treatment group will be presented by MedDRA system organ class, preferred term, and treatment group in Table 57.
- The number of subjects reporting adverse events occurring in 5% of subjects in any treatment group presented by MedDRA system organ class, preferred term and treatment group in Table 57.
- Subject listing of non-serious adverse events of moderate or greater severity (Table 58);
- Bar chart of total frequency of adverse events by severity and MedDRA system organ class (Figure 4);
- Bar chart of subject incidence of adverse events by severity and MedDRA system organ class (Figure 5);

#### 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

A listing of deaths and serious adverse events will be presented, which will include Subject ID, treatment group, Adverse Event Description, Study Day the Event became Serious, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if Not Related, Outcome, and Duration of Event in days (Table 59).

# 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of the total pregnancies, number of live births, and number of spontaneous abortions, elective abortions or still births will be presented (Listing 21, Listing 22, Listing 23, Listing 24, and Listing 25).

### 9.6. Clinical Laboratory Evaluations

Several clinical laboratory parameters are collected at screening and Visit 2. The evaluations are: urine pregnancy test, vaginal swab specimens for NAAT testing for trichomonas, quantitative NAAT testing for GV and NAAT testing for *T. vaginalis*, a vaginal swab specimen to determine the vaginal pH using ColorpHast pH paper, and a vaginal swab for microbiologic assessment of BV by Nugent criteria.

Individual clinical laboratory results will be provided in Listing 6 for all enrolled subjects and Listing 7 for subjects who were GV negative at baseline.

# 9.7. Vital Signs and Physical Evaluations

A pelvic examination will be performed at screening and Visit 2 for the collection of vaginal swab specimens for: pH, whiff test, and wet prep microscopy (Amsel criteria with the exception of evaluation of vaginal discharge), Nugent score, NAAT for trichomonas, quantitative NAAT for GV, and future use. A subject listing will be provided for all findings (Listing 26). Other gynecological test results including KOH saline microscopy will be presented in Listing 27 and BV microbiology results will be presented in Listing 28.

# 10. PHARMACOKINETICS

Not applicable for this study.

# 11. IMMUNOGENICITY

Not applicable for this study.

# 12. OTHER ANALYSES

There are no additional analyses planned for this study.

#### 13. REPORTING CONVENTIONS

P-values  $\ge$ 0.001 and  $\le$ 0.999 will be reported to three decimal places; p-values less than 0.001 will be reported as "<0.001"; p-values greater than 0.999 will be reported as ">0.999". The mean, median, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles other than the median will use the same number of decimal places as the original data. Proportions will be presented to two decimal places; values <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values <1% will be presented as "<1". Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to three significant figures.

# 14. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

# 16. REFERENCES

1. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.

# 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3, respectively.
## **APPENDICES**

## APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Study Design | 35 |
|---|---|---|
| Table 2: | Schedule of Study Procedures | 37 |
| Table 3: | Dates of First Treatment by Site – Safety Population | 38 |
| Table 4: | Dates of First Treatment by Treatment Group - Safety Population | 39 |
| Table 5: | Safety and Per-Protocol Analysis Population Eligibilities for Safety and Primary Efficacy Analysis by Treatment Group | 40 |
| Table 6: | Summary of Halting Rules - Safety Population | 41 |
| Table 7: | Ineligibility Summary of Screen Failures | 42 |
| Table 8: | Subject Disposition by Treatment Group - All Enrolled Subjects | 43 |
| Table 9: | Distribution of Protocol Deviations by Category, Type, and Treatment<br>Group - All Enrolled Subjects | 44 |
| Table 10: | GV Eradication at Visit 2 by Treatment Group - ITT Population | 46 |
| Table 11: | GV Eradication at Visit 2 by Treatment Group - PP Population | 46 |
| Table 12: | Summary of Amsel Criteria by Treatment Group and Study Visit – ITT Population | 47 |
| Table 13: | Summary of Amsel Criteria by Treatment Group and Study Visit – PP Population | 47 |
| Table 14: | Amsel Criteria at Visit 2 by GV Eradication Status and Treatment Group - ITT Population | 48 |
| Table 15: | Amsel Criteria at Visit 2 by GV Eradication Status and Treatment Group - PP Population | 48 |
| Table 16: | Nugent Scores by Category, Study Visit, and Treatment Group - ITT Population | 49 |
| Table 17: | Nugent Scores by Category, Study Visit, and Treatment Group - PP Population | 49 |
| Table 18: | Continuous Nugent Score Characteristics by Study Visit, and Treatment Group - ITT Population | 50 |
| Table 19: | Continuous Nugent Score Characteristics by Study Visit, and Treatment Group - PP Population | 50 |
| Table 20: | Nugent Scores at Visit 2 by Category, GV Eradication Status, and Treatment Group - ITT Population | 51 |
| Table 21: | Nugent Scores at Visit 2 by Category, GV Eradication Status, and Treatment Group - PP Population | 51 |

| Table 22: | Continuous Nugent Score Characteristics at Visit 2 by GV Eradication Status and Treatment Group - ITT Population | 52 |
|---|---|---|
| Table 23: | Continuous Nugent Score Characteristics at Visit 2 by GV Eradication Status and Treatment Group - PP Population | 52 |
| Table 24: | Mean count of <i>Lactobacillus spp.</i> , <i>Gardnerella/Bacteroides spp.</i> , and <i>Mobiluncus spp.</i> By Study Visit, and Treatment Group – ITT Population | 53 |
| Table 25: | Mean count of <i>Lactobacillus spp.</i> , <i>Gardnerella/Bacteroides spp.</i> , and <i>Mobiluncus spp.</i> by Study Visit, and Treatment Group - PP Population | 53 |
| Table 26: | Mean count of <i>Lactobacillus spp.</i> , <i>Gardnerella/Bacteroides spp.</i> , and <i>Mobiluncus spp.</i> At Visit 2 by GV Eradication Status and Treatment Group - ITT Population | 54 |
| Table 27: | Mean count of <i>Lactobacillus spp.</i> , <i>Gardnerella/Bacteroides spp.</i> , and <i>Mobiluncus spp.</i> At Visit 2 by GV Eradication Status and Treatment Group - PP Population | 54 |
| Table 28: | Summary of Categorical Demographic and Baseline Characteristics by GV<br>Status at Screening - NAAT Screening Population | 55 |
| Table 29: | Summary of Continuous Demographic and Baseline Characteristics by GV Status at Screening – NAAT Screening Population | 56 |
| Table 30: | Categorical Baseline Sexual History by GV Status at Screening - NAAT Screening Population | 57 |
| Table 31: | Continuous Baseline Sexual History by GV Status at Screening – NAAT Screening Population | 58 |
| Table 32: | Categorical Baseline Sexual History by Visit 2 BV Status - ITT Population – Amoxicillin Treatment Group | 60 |
| Table 33: | Categorical Baseline Sexual History by Visit 2 BV Status - ITT Population – Placebo Treatment Group | 61 |
| Table 34: | Continuous Baseline Sexual History by Visit 2 BV Status - ITT Population – Amoxicillin Treatment Group | 62 |
| Table 35: | Continuous Baseline Sexual History by Visit 2 BV Status - ITT Population – Placebo Treatment Group | 63 |
| Table 36: | Summary of Categorical Demographic and Baseline Characteristics by Visit 2 BV Status - ITT Population – Amoxicillin Treatment Group | 64 |
| Table 37: | Summary of Categorical Demographic and Baseline Characteristics by Visit 2 BV Status - ITT Population – Placebo Treatment Group | 64 |
| Table 38: | Summary of Continuous Demographic and Baseline Characteristics by Visit 2 BV Status – ITT Population – Amoxicillin Treatment Group | 65 |
| Table 39: | Summary of Continuous Demographic and Baseline Characteristics by Visit 2 BV Status – ITT Population – Placebo Treatment Group | |

| Table 40: | Summary of Categorical Demographic and Baseline Characteristics by Site - All Enrolled Subjects | 66 |
|---|---|---|
| Table 41: | Summary of Categorical Demographic and Baseline Characteristics by<br>Treatment Group - ITT Population | 67 |
| Table 42: | Summary of Continuous Demographic and Baseline Characteristics by Site—All Enrolled Subjects. | 68 |
| Table 43: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group - ITT Population | 69 |
| Table 44: | Categorical Baseline Sexual History by Treatment Group -ITT Population | 70 |
| Table 45: | Continuous Baseline Sexual History by Treatment Group-ITT Population | 71 |
| Table 46: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population – All Sites | 73 |
| Table 47: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population – University of Alabama at Birmingham | 73 |
| Table 48: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population – Wake Forest University Health Sciences | 73 |
| Table 49: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - All Subjects | 74 |
| Table 50: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - University of Alabama at Birmingham | 74 |
| Table 51: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - Wake Forest University Health Sciences | 74 |
| Table 52: | Proportion of Subjects Reporting Treatment Related Adverse Events Following the First Dose of Treatment through Visit 2 by Treatment Group – Safety Population | 75 |
| Table 53: | Proportion of Subjects Discontinuing Treatment Early Due to Adverse Events by Treatment Group – Safety Population | 76 |
| Table 54: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population | 77 |
| Table 55: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity and Relationship - Safety Population | 78 |

| Table 56: | Number and Percentage of Subjects Experiencing Unsolicited Adverse<br>Events by MedDRA System Organ Class and Preferred Term, Maximum<br>Severity, Relationship, and Treatment Group - Safety Population | 79 |
|---|---|---|
| Table 57: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class, Preferred Term, and Treatment Group - Safety Population | 80 |
| Table 58: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 81 |
| Table 59: | Listing of Serious Adverse Events | 82 |

**Table 1:** Study Design

Study Visit 0: Screening

Total N: ~245 screened to enroll 98 (to achieve 82 evaluable)

Screening: obtain informed consent; perform screening; collect demographics, sexual history, medical history and concomitant medications; conduct clinical assessments and pregnancy test

Samples Collected: Urine for pregnancy testing; Vaginal swab specimen for testing of

Samples Collected: Urine for pregnancy testing; Vaginal swab specimen for testing of yeast, trichomonas and BV/abnormal vaginal flora and NAAT testing for T. vaginalis; Vaginal swab specimen for testing of GV, BV, and future use



## Study Visit 1: Enrollment

Enrollment: review tests results from Screening Visit, review eligibility, obtain informed consent; collect interim sexual history, medical history, and concomitant medications



Dispense study product and issue participant memory aid

Remind all participants to abstain from vaginal intercourse or use a condom to prevent

GV reinfection



Study Visit 2: Follow-up (ToC) Collect interim sexual history, medical history, and concomitant medications; assess AEs;

#### conduct clinical assessment

Samples Collected: Vaginal swab specimen for testing of yeast, trichomonas and BV/abnormal vaginal flora; Vaginal swab specimen for testing of GV, BV, and future use



**Table 2:** Schedule of Study Procedures

| | | Screening | Enrollment | Follow-Up | pa | u |
|---|---|---|---|---|---|---|
| | | Visit 0<br>(Day -14 to -7) | Visit 1<br>(Day 1) | Visit 2<br>(Day 15<br>[Window: 15-21]) | Unscheduled | Early<br>Termination |
| Signed Consent Form <sup>1</sup> | | X | X | | | |
| Assessment of Eligibility | y Criteria | X | X | | | |
| Collection of Demograp | hics | X | | | | |
| Review of Sexual Histor | у | X | X | X | (X) | X |
| Review of Medical Histo | ory <sup>2</sup> | X | X | X | (X) | X |
| Review of Concomitant | Medications | X | X | X | (X) | X |
| Randomization | | | X | | | |
| Dispense memory aid an | nd instructions | | X | | | |
| Reminder on abstinence to prevent GV reinfectio | Reminder on abstinence or condom use during vaginal intercourse to prevent GV reinfection | | X | | | |
| Study Intervention | | | X | | | |
| Pelvic Examination | | X | | X | (X) | (X) |
| Assessment of Adverse | Events | | | X | X | X |
| Assessment of study dru and drug return) | g compliance (via review of memory aid | | | X | (X) | (X) |
| | Urine Pregnancy Test | X | | | | |
| Clinical Laboratory | Trichomonas, NAAT Test | X | | | | |
| | pH, whiff test, and wet microscopy (Amsel criteria) | X | | X | (X) | (X) |
| Research Laboratory | BV, Nugent score | X | | X | (X) | (X) |
| Research Laboratory | Future Use <sup>3</sup> | X | | X | (X) | (X) |
| LabCorp | GV, quantitative NAAT | X | | X | (X) | (X) |

<sup>(</sup>X) – As indicated/appropriate.

At Visit 0 the participant is signing the Screening Informed Consent Form. At Visit 1 the participant will then sign the Enrollment Informed Consent Form.

<sup>&</sup>lt;sup>2</sup> Medical history is to be originally collected only on active conditions within one year prior to screening. Then at follow up visits, the active conditions will be reviewed and any new conditions captured.

<sup>&</sup>lt;sup>3</sup> At Visit 0 Screening and at Visit 2, participants that agree will have an extra swab specimen collected for future use.

**Table 3:** Dates of First Treatment by Site – Safety Population

[Note: Dates will be categorized by breaking the calendar year into quarters.]

| Dates of Dosing | University of Alabama at Birmingham (N = X) | | Scie | niversity Health<br>ences<br>= X) | All Subjects (N = X) | |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| DDMMMYYYY-<br>DDMMMYYYY | X | X | X | X | Х | Х |
| DDMMMYYYY-<br>DDMMMYYYY | X | X | Х | X | Х | Х |
| DDMMMYYYY-<br>DDMMMYYYY | X | X | X | X | Х | X |
| DDMMMYYYY-<br>DDMMMYYYY | X | X | X | X | Х | X |

N=Number of subjects in the safety population of each site.

**Table 4:** Dates of First Treatment by Treatment Group - Safety Population

[Implementation Note: Dates will be categorized by breaking the calendar year into quarters.]

| Dates of Dosing | Amoxicillin<br>(N = X) | | | Placebo<br>(N = X) | All Subjects (N = X) | |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | X | X |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | X | X |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | Х | X |
| DDMMMYYYY-DDMMMYYYY | X | X | X | X | х | X |

N=Number of subjects in the safety population who received the specified treatment group. Treatment group is the actual treatment received.

Table 5: Safety and Per-Protocol Analysis Population Eligibilities for Safety and Primary Efficacy Analysis by Treatment Group

| | | | | xicillin<br>=X) | Placebo<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|
| Analysis Population | Eligibility Category | Reason Subjects Excluded | n | % | n | % | n | % |
| | Eligible for Safety | | X | х | х | х | х | X |
| Safety Analysis Population | F1-1-1-1-1 | Any Reason | X | х | х | х | х | X |
| | Excluded from Safety | Did not receive study product | X | х | х | х | х | X |
| | Eligible for PP | | X | х | х | х | х | X |
| | | Any Reason | х | х | х | х | х | x |
| | | Did not meet inclusion/exclusion criteria | X | x | х | х | х | x |
| | | Was not evaluable | X | x | х | х | х | x |
| Per-Protocol (PP) Analysis | | Did not use 80% of the scheduled doses | X | x | х | х | х | x |
| Population | Excluded from PP | Did not return for the Test of Cure Visit within window (Day 15-21) | x | x | х | x | x | x |
| | | Unprotected vaginal sexual intercourse between Visit 1 and Visit 2 | X | x | х | x | x | X |
| | | Pregnancy reported | X | x | х | x | x | X |
| | | Received an antibiotic or intravaginal microbicide other than study drug | Х | х | х | х | х | Х |

N=Number of subjects enrolled in the specified treatment group.

Treatment group is the actual treatment a subject received

## **Table 6:** Summary of Halting Rules - Safety Population

| Halting Rules | Number of<br>Subjects |
|---|---|
| Two participants experience an adverse event that is judged to be Severe (Grade 3) and related to study product | X |

**Table 7:** Ineligibility Summary of Screen Failures

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | Number of Subjects <sup>a</sup> |
|---|---|---|
| Inclusion and Exclusion | Any Criterion | x |
| Inclusion | Any inclusion criterion | x |
| | [inclusion criterion 1] | x |
| | [inclusion criterion 2] | x |
| | [inclusion criterion 3] | x |
| Exclusion | Any exclusion criterion | x |
| | [exclusion criterion 1] | x |
| | [exclusion criterion 2] | x |
| | [exclusion criterion 3] | x |
| Declined Enrollment | Any Reason | x |
| | Time commitment | x |
| | Concern of potential risks | x |
| | Number of procedures | x |
| | Unable to contact subject | x |
| | Other | x |

<sup>&</sup>lt;sup>a</sup>More than one criterion may be marked per subject.

Table 8: **Subject Disposition by Treatment Group - All Enrolled Subjects** 

| Subject | Amoxicillin<br>(N=X) | | | cebo<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|
| Disposition | n | % | n | % | n | % |
| Screened | | | | | X | |
| Evaluated for GV via NAAT | X | X | X | X | X | X |
| GV Negative <sup>1</sup> | X | X | X | X | х | Х |
| GV Positive* | X | X | X | X | х | Х |
| Enrolled/Randomized | X | 100 | X | 100 | х | 100 |
| Received Treatment | X | X | X | X | х | Х |
| Complied with Treatment <sup>2,3</sup> | х | X | X | X | х | Х |
| Completed Visit 2 (Day 15-21) | х | X | X | X | х | X |

N=Number of subjects who received the specified treatment.

Treatment group is the treatment to which the subject was randomized.

<sup>1</sup>The denominators for the percentages is the number of subjects evaluated for GV.

<sup>2</sup>Refer to Listing 3 for reasons subjects discontinued or terminated early.

<sup>3</sup>Refer to Listing 15 and 16 for treatment compliance.

 Table 9:
 Distribution of Protocol Deviations by Category, Type, and Treatment Group - All Enrolled Subjects

| | | | moxicill<br>(N=X) | in | Placebo<br>(N=X) | | | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. |
| Eligibility/enrollment | Any type | X | Х | х | x | Х | X | Х | X | х |
| | Did not meet inclusion criterion | х | х | х | х | х | Х | х | х | х |
| | Met exclusion criterion | x | X | х | X | X | X | X | X | X |
| | ICF not signed prior to study procedures | X | х | х | X | х | X | Х | х | х |
| | Other | X | х | х | X | х | X | Х | х | х |
| Treatment administration schedule | Any type | X | х | х | X | х | X | Х | х | х |
| | Out of window visit | X | х | х | X | х | X | Х | х | х |
| | Other | х | X | х | x | х | X | х | Х | х |
| Follow-up visit schedule | Any type | х | X | х | x | х | X | х | Х | х |
| | Out of window visit | х | Х | х | x | х | x | х | х | x |
| | Missed visit/visit not conducted | х | Х | х | x | х | x | х | х | x |
| | Other | х | Х | х | x | х | x | х | х | x |
| Protocol procedure/assessment | Any type | x | Х | х | х | х | X | х | х | x |
| | Incorrect version of ICF signed | x | Х | х | х | х | X | х | х | x |
| | Blood not collected | х | Х | х | х | х | х | X | х | х |
| | Urine not collected | х | Х | х | х | х | х | X | х | х |
| | Other specimen not collected | х | Х | х | х | х | х | X | х | х |
| | Specimen result not obtained | х | Х | х | х | х | х | х | х | х |
| | Required procedure not conducted | X | х | х | х | х | x | х | х | x |
| | Required procedure done incorrectly | X | х | х | х | х | x | х | х | x |
| | Study product temperature excursion | X | х | х | х | х | x | х | х | x |
| | Specimen temperature excursion | X | х | х | х | х | x | х | х | x |
| | Prohibited use of vaginal products | х | х | х | X | х | X | X | х | Х |

Table 9: Distribution of Protocol Deviations by Category, Type, and Treatment Group - All Enrolled Subjects (Continued)

| | | | noxicilli<br>(N=X) | in | | Placebo<br>(N=X) | | | l Subjec<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. | # of<br>Subj. | % | # of<br>Dev. |
| | Other | х | x | x | х | х | Х | X | X | x |
| Treatment administration | Any type | х | X | X | x | X | X | X | X | X |
| | Required procedure done incorrectly | х | X | X | х | х | Х | X | X | х |
| | Study product temperature excursion | х | х | х | х | х | Х | X | X | х |
| | Other | х | X | X | х | х | Х | X | X | х |
| Blinding policy/procedure | Any type | х | X | X | х | х | Х | X | X | х |
| | Treatment unblinded | х | х | х | х | х | Х | х | X | х |
| | Other | x | х | х | х | х | х | Х | х | Х |

N=Number of subjects who received the specified treatment. Treatment group is the treatment to which the subject was randomized.

Implementation Note: Only include the Deviation Types that are reported in the study, i.e. delete any rows with # of Dev = 0.

Table 10: GV Eradication at Visit 2 by Treatment Group - ITT Population

| Imputation<br>Method | Treatment<br>Group | Number of<br>Subjects with<br>GV Eradication<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with GV<br>Eradication | Proportion of<br>Subjects with GV<br>Eradication<br>95% CI <sup>1</sup> | Difference in Proportion of<br>Subjects with GV<br>Eradication between<br>Amoxicillin and Placebo | Difference in Proportion of<br>Subjects with GV Eradication<br>between Amoxicillin and Placebo<br>95% CI | P-Value <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| | Amoxicillin | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| ITT Treatment Failure | Placebo | X | X | 0.xx | 0.xx, 0.xx | | | |
| Tandie | All Subjects | X | x | 0.xx | 0.xx, 0.xx | | | |
| | Amoxicillin | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| ITT Worst Case<br>Imputation | Placebo | X | х | 0.xx | 0.xx, 0.xx | | | |
| imputation | All Subjects | X | х | 0.xx | 0.xx, 0.xx | | | |

The denominator for proportions is based on the number of subjects who received the specified treatment and analysis population.

Tables with similar format:

## Table 11: GV Eradication at Visit 2 by Treatment Group - PP Population

Implementation Note: Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received."

Treatment group is the treatment to which the subject was randomized.

<sup>&</sup>lt;sup>1</sup>95% CI = 95% Wilson confidence interval.

<sup>&</sup>lt;sup>2</sup>P-value from the two-sided Pearson Chi-Square test with Yates continuity correction at the .05 level of significance.

Table 12: Summary of Amsel Criteria by Treatment Group and Study Visit – ITT Population

| | | | | xicillin<br>=X) | | | | cebo<br>=X) | | | | bjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Amsel Criteria | | Scree<br>(N= | | | sit 2<br>=X) | | ening<br>=X) | Vis<br>(N= | sit 2<br>=X) | Scree<br>(N= | ening<br>=X) | | sit 2<br>=X) |
| | | n | % | n | % | n | % | n | % | n | % | n | % |
| | 0/3 | X | Х | x | x | X | X | X | X | X | X | x | Х |
| Number of Amsel Criteria | 1/3 | X | X | X | x | X | X | x | X | X | X | X | X |
| Present | 2/3 | Х | Х | х | х | х | X | х | X | X | Х | х | х |
| | 3/3 | X | Х | x | x | X | X | X | X | X | X | x | Х |
| 37 ' 1 II | >4.5 | Х | Х | х | х | х | X | х | X | X | Х | х | х |
| Vaginal pH | ≤4.5 | Х | Х | х | х | х | X | х | X | X | Х | х | х |
| Cl. C. II | ≥20% | х | х | х | х | х | х | х | x | X | Х | х | Х |
| Clue Cells | <20% | х | х | X | х | X | X | x | X | X | Х | x | х |
| WILCOT A | Positive | х | х | X | х | X | X | x | X | X | Х | x | х |
| Whiff Test | Negative | X | X | X | х | х | Х | х | х | X | X | х | X |

Denominator for percentages is the number of subjects who received the specified treatment.

Treatment group is the treatment to which the subject was randomized.

#### Tables with similar format:

## Table 13: Summary of Amsel Criteria by Treatment Group and Study Visit – PP Population

Implementation Note: Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received"

Table 14: Amsel Criteria at Visit 2 by GV Eradication Status and Treatment Group - ITT Population

| | | | | | xicillin<br>(=X) | | | | | | icebo<br>i=X) | | | | | | ubjects<br>=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Amsel Criteria | | Erac | GV<br>licated<br>I=X) | Era | V Not<br>dicated<br>N=X) | Eva | Not<br>luable<br>(=X) | Erac | GV<br>licated<br>I=X) | Era | V Not<br>dicated<br>N=X) | Eva | Not<br>luable<br>V=X) | Erac | GV<br>dicated<br>V=X) | Erac | Not<br>licated<br>(=X) | Eval | lot<br> uable<br> =X) |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | 0/3 | X | X | X | х | X | X | X | X | X | х | Х | Х | Х | Х | X | X | X | X |
| Number of Amsel | 1/3 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Criteria Present | 2/3 | X | X | X | х | Х | X | X | X | X | х | X | Х | Х | Х | X | X | X | X |
| | 3/3 | X | X | X | х | Х | X | X | X | X | х | X | Х | Х | Х | X | X | X | X |
| Vacinal all | >4.5 | X | X | X | х | Х | X | X | X | X | х | X | Х | Х | Х | X | X | X | X |
| Vaginal pH | ≤4.5 | X | X | X | х | Х | X | X | X | X | х | X | Х | Х | Х | X | X | X | X |
| Class Calla | ≥20% | X | X | X | х | X | X | X | X | X | х | X | X | Х | X | X | X | X | X |
| Clue Cells | <20% | X | X | х | х | Х | X | х | х | х | х | х | Х | Х | Х | X | х | Х | X |
| WILLIES T | Positive | х | Х | Х | х | х | х | х | х | Х | х | х | х | х | Х | х | х | х | X |
| Whiff Test | Negative | Х | X | X | Х | Х | х | х | X | X | х | х | Х | х | х | X | X | Х | Х |

Denominator for percentages is the number of subjects who received the specified treatment.

Treatment group is the treatment to which the subject was randomized.

#### Tables with Similar Format:

## Table 15: Amsel Criteria at Visit 2 by GV Eradication Status and Treatment Group - PP Population

#### Implementation Note:

- 1. Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received."
- 2. No "Not Evaluable" Column for PP Population.

Table 16: Nugent Scores by Category, Study Visit, and Treatment Group - ITT Population

| | | | xicillin<br>=X) | | | | cebo<br>=X) | | | | ıbjects<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screeni<br>(N = | ng Visit<br>= X) | | sit 2<br>= X) | Screeni<br>(N = | ng Visit<br>= X) | | it 2<br>= X) | Screeni<br>(N = | ng Visit<br>= X) | Vis<br>(N = | it 2<br>= X) |
| | n | % | n | % | n | % | n | % | n | % | n | % |
| 0-3 (Normal) | Х | X | х | х | Х | X | X | X | х | Х | X | х |
| 4-6 (Intermediate) | X | X | X | Х | X | X | X | X | X | X | X | Х |
| 7-10 (BV) | Х | X | х | х | Х | X | X | X | х | Х | X | х |

Denominator for percentages is the number of subjects who received the specified treatment.

Treatment group is the treatment to which the subject was randomized.

Tables with similar format:

## Table 17: Nugent Scores by Category, Study Visit, and Treatment Group - PP Population

Implementation Note: Change footnote from "Treatment group is the treatment to which the subject was randomized." To "Treatment group is the actual treatment received."

Table 18: Continuous Nugent Score Characteristics by Study Visit, and Treatment Group - ITT Population

| | | icillin<br>=X) | Plac<br>(N= | eebo<br>=X) | All Su<br>(N= | • |
|---|---|---|---|---|---|---|
| Statistic | Screening Visit (N = X) | Visit 2<br>(N = X) | Screening Visit (N = X) | Visit 2<br>(N = X) | Screening Visit (N = X) | Visit 2<br>(N = X) |
| Mean | x.x | x.x | x.x | x.x | x.x | x.x |
| Standard Deviation of Mean | x.x | x.x | x.x | x.x | x.x | x.x |
| Mean Change from Visit 1 | | x.x | | x.x | | x.x |
| Standard Deviation of Mean Change from Visit 1 | | x.x | | x.x | | x.x |

Treatment group is the treatment to which the subject was randomized.

Tables with similar format:

## Table 19: Continuous Nugent Score Characteristics by Study Visit, and Treatment Group - PP Population

Implementation Note: Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received."

Table 20: Nugent Scores at Visit 2 by Category, GV Eradication Status, and Treatment Group - ITT Population

| | | | | noxicillin<br>(N=X) | | | Placebo<br>(N=X) | | | | | | | | Subjects<br>N = X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nugent Score<br>Category | Erad | GV<br>licated<br>= X) | Erac | V Not<br>licated<br>= X) | | valuable<br>= X) | Erac | GV<br>licated<br>= X) | Erac | Not licated = X) | | valuable<br>= X) | Erac | GV<br>licated<br>= X) | Erac | Not<br>licated<br>= X) | | valuable<br>= X) |
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| 0-3 (Normal) | х | X | X | X | X | x | X | X | х | X | X | X | X | X | X | X | X | x |
| 4-6 (Intermediate) | х | X | х | Х | Х | х | х | Х | х | Х | Х | X | х | X | X | X | X | х |
| 7-10 (BV) | х | х | х | х | х | х | Х | Х | х | х | х | х | х | X | Х | X | X | х |

Denominator for percentages is the number of subjects in the ITT population for each treatment group.

Treatment group is the treatment to which the subject was randomized.

#### Tables with similar format:

## Table 21: Nugent Scores at Visit 2 by Category, GV Eradication Status, and Treatment Group - PP Population

## Implementation Note:

- 1. Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received.
- 2. No "Not Evaluable" Column for PP Population.

Table 22: Continuous Nugent Score Characteristics at Visit 2 by GV Eradication Status and Treatment Group - ITT Population

| | | Amoxicillin<br>(N=X) | | | Placebo<br>(N=X) | | | All Subjects (N = X) | |
|---|---|---|---|---|---|---|---|---|---|
| Statistic | GV<br>Eradicated<br>(N = X) | GV Not<br>Eradicated<br>(N = X) | Not<br>Evaluable<br>(N = X) | GV<br>Eradicated<br>(N = X) | GV Not<br>Eradicated<br>(N = X) | Not<br>Evaluable<br>(N = X) | GV<br>Eradicated<br>(N = X) | GV Not<br>Eradicated<br>(N = X) | Not<br>Evaluable<br>(N = X) |
| Mean | x.x | x.x | X.X | x.x | x.x | x.x | x.x | x.x | X.X |
| Standard Deviation of Mean | X.X | X.X | X.X | X.X | x.x | X.X | X.X | X.X | X.X |
| Mean Change from Visit 1 | X.X | X.X | X.X | X.X | x.x | X.X | X.X | X.X | X.X |
| Standard Deviation of Mean<br>Change from Visit 1 | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |

Treatment group is the treatment to which the subject was randomized.

#### Tables with similar format:

## Table 23: Continuous Nugent Score Characteristics at Visit 2 by GV Eradication Status and Treatment Group - PP Population

## Implementation Note:

- 1. Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received."
- 2. No "Not Evaluable" Column for PP Population.

Table 24: Mean count of *Lactobacillus spp.*, *Gardnerella/Bacteroides spp.*, and *Mobiluncus spp.* By Study Visit, and Treatment Group – ITT Population

| | | - | xicillin<br>=X) | Plac<br>(N= | eebo<br>=X) | | bjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Species | Statistic | Screening<br>Visit<br>(N = X) | Visit 2<br>(N = X) | Screening<br>Visit<br>(N = X) | Visit 2<br>(N = X) | Screening<br>Visit<br>(N = X) | Visit 2<br>(N = X) |
| | Mean | x.x | X.X | X.X | X.X | X.X | x.x |
| I gotob goillug gnn | Standard Deviation of Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| Lactobacillus spp. | Mean Change from Screening | | X.X | | X.X | | X.X |
| | Standard Deviation of Mean Change from Screening | | X.X | | X.X | | X.X |
| | Mean | X.X | X.X | X.X | X.X | x.x | X.X |
| Conducatella/Doctorida | Standard Deviation of Mean | X.X | X.X | X.X | X.X | x.x | X.X |
| Gardnerella/Bacteroides spp | Mean Change from Screening | | X.X | | X.X | | X.X |
| | Standard Deviation of Mean Change from Screening | | X.X | | X.X | | X.X |
| | Mean | X.X | X.X | X.X | X.X | x.x | X.X |
| Mahilungua ann | Standard Deviation of Mean | X.X | X.X | x.x | x.x | x.x | X.X |
| Mobiluncus spp | Mean Change from Screening | | X.X | | x.x | | X.X |
| | Standard Deviation of Mean Change from Screening | | X.X | | X.X | | X.X |

Treatment group is the treatment to which the subject was randomized.

Tables with similar format:

# Table 25: Mean count of *Lactobacillus spp.*, *Gardnerella/Bacteroides spp.*, and *Mobiluncus spp.* by Study Visit, and Treatment Group - PP Population

Implementation Note: Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received."

Table 26: Mean count of *Lactobacillus spp.*, *Gardnerella/Bacteroides spp.*, and *Mobiluncus spp.* At Visit 2 by GV Eradication Status and Treatment Group - ITT Population

| | | | Amoxicillin (N=X) | | | Placebo<br>(N=X) | | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Species | Statistic | GV<br>Eradicated<br>(N = X) | GV Not<br>Eradicated<br>(N = X) | Not<br>Evaluable<br>(N = X) | GV<br>Eradicated<br>(N = X) | GV Not<br>Eradicated<br>(N = X) | Not<br>Evaluable<br>(N = X) | GV<br>Eradicated<br>(N = X) | GV Not<br>Eradicated<br>(N = X) | Not<br>Evaluable<br>(N = X) |
| Lactobacillus spp. | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Laciovaciius spp. | Standard Deviation of Mean | X.X | x.x | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Gardnerella/Bacteroides | Mean | X.X | x.x | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| spp | Standard Deviation of Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| Makikanana | Mean | x.x | x.x | x.x | x.x | X.X | x.x | x.x | x.x | X.X |
| Mobiluncus spp | Standard Deviation of Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |

Treatment group is the treatment to which the subject was randomized.

## Tables with similar format:

Table 27: Mean count of *Lactobacillus spp.*, *Gardnerella/Bacteroides spp.*, and *Mobiluncus spp.* At Visit 2 by GV Eradication Status and Treatment Group - PP Population

## Implementation Note:

- 1. Change footnote from "Treatment group is the treatment to which the subject was randomized." to "Treatment group is the actual treatment received."
- 2. No "Not Evaluable" Column for PP Population.

Table 28: Summary of Categorical Demographic and Baseline Characteristics by GV Status at Screening - NAAT Screening Population

| | | | ositive<br>=X) | GV Neg<br>(N=2 | |
|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % |
| Sex | Female | х | xx | X | xx |
| Ethnicity | Not Hispanic or Latino | х | xx | X | xx |
| | Hispanic or Latino | х | xx | X | xx |
| | Not Reported | х | xx | X | xx |
| | Unknown | х | xx | X | xx |
| Race | American Indian or Alaska Native | х | xx | X | xx |
| | Asian | х | xx | X | xx |
| | Native Hawaiian or Other Pacific Islander | х | xx | X | xx |
| | Black or African American | х | xx | X | xx |
| | White | х | xx | X | xx |
| | Multi-Racial | х | XX | X | xx |
| | Unknown | х | XX | X | xx |

N=Number of Subjects in the GV NAAT population within the specified GV status category.

Table 29: Summary of Continuous Demographic and Baseline Characteristics by GV Status at Screening – NAAT Screening Population

| Variable | Statistic | GV Positive<br>(N=X) | GV Negative<br>(N=X) |
|----------|--------------------|----------------------|----------------------|
| Age | Mean | X.X | X.X |
| | Standard Deviation | X.X | X.X |
| | Median | X.X | X.X |
| | Minimum | X | X |
| | Maximum | X | X |

N=Number of Subjects in the GV NAAT population within the specified GV status category.

Table 30: Categorical Baseline Sexual History by GV Status at Screening - NAAT Screening Population

| Sexual Behavior Category | Value | GV Pos<br>(N=2 | | GV Negative<br>(N=X) | |
|---|---|---|---|---|---|
| | | n | % | n | % |
| Has the subject ever douched or used vaginal preparations or drying agents? | No | X | x | X | X |
| | Summer's Eve | X | x | X | X |
| | Rephresh | X | x | X | X |
| | Vagisil | X | x | X | X |
| | Other | X | x | X | X |
| Does the subjects have a history of recurrent BV (more than one episode | No | X | x | X | X |
| of BV in the prior 12 months)? | Yes | X | x | X | X |
| Did the subject have a diagnosis of BV within the prior 6 months? | No | X | x | X | X |
| Did the subject have a diagnosis of BV within the prior 6 months: | Yes | X | x | X | X |
| | Was a new partner | X | X | X | X |
| Subject's most recent sexual partner | Was a male | X | x | X | X |
| Subject's most recent sexual partner | Used a condom | X | x | X | X |
| | N/A | X | x | X | X |
| In the last 30 days, how often did the subject use a condom? | Always | X | X | X | X |
| | Sometimes | X | x | X | X |
| | Never | х | x | X | X |
| In the last 3 months, how often did the subject use a condom? | Always | х | x | X | X |
| | Sometimes | X | x | X | X |
| | Never | X | X | X | X |

N=Number of Subjects in the GV NAAT population within the specified GV status category.

Screening Visit 0.

Denominator for percentages is the number of subjects screened with male partners in the specified time frame.

Table 31: Continuous Baseline Sexual History by GV Status at Screening – NAAT Screening Population

| Time Frame | Sexual Behavior Characteristic | Statistic | Baseline GV Positive (N=X) | Baseline GV Negative<br>(N=X) |
|---|---|---|---|---|
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Days since the subject last had sexual intercourse | Median | x.x | X.X |
| | intercourse | Minimum, Maximum | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of episodes of BV in prior 12 months | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | X, X |
| | Number of times the subject douched | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | or used vaginal preparations or drying | Median | x.x | X.X |
| | agents | Minimum, Maximum | x, x | X, X |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Total number of partners | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | X, X |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of new partners | Median | x.x | X.X |
| In the last 30 days | | Minimum, Maximum | x, x | X, X |
| in the last 30 days | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of regular partners | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | X, X |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of occasional partners | Median | X.X | X.X |
| | | Minimum, Maximum | X, X | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of male partners | Median | X.X | X.X |
| | | Minimum, Maximum | x, x | X, X |

Table 31: Continuous Baseline Sexual History by GV Status at Screening – NAAT Screening Population (Continued)

| Time Frame | Sexual Behavior Characteristic | Statistic | Baseline GV Positive<br>(N=X) | Baseline GV Negative<br>(N=X) |
|---|---|---|---|---|
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Total number of partners | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | X, X |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of new partners | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| In the last 3 months | Number of regular partners | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of occasional partners | Median | x.x | X.X |
| | | Minimum, Maximum | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) |
| | Number of male partners | Median | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x |

N = Number of subjects in the NAAT Screening Population within the specified GV status category. Screening Visit 0.

Table 32: Categorical Baseline Sexual History by Visit 2 BV Status - ITT Population – Amoxicillin Treatment Group

| | | | Amoxicil | lin (N=X) | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Sexual Behavior Category | Value | BV by Amsel Criteria<br>(N=X) | | BV by Nugent Score<br>(N=X) | | BV by Amsel Criteria and<br>Nugent Score<br>(N=X) | | No BV by either Amsel or<br>Nugent Score<br>(N=X) | |
| | | n | % | n | % | n | % | n | % |
| Has the subject ever douched or used vaginal | No | х | X | х | х | Х | x | x | х |
| preparations or drying agents? | Summer's Eve | x | X | X | Х | X | x | x | X |
| | Rephresh | X | X | х | х | X | x | x | X |
| | Vagisil | х | X | х | х | X | x | x | Х |
| | Other | х | X | х | х | X | x | x | Х |
| Does the subjects have a history of recurrent BV (more than one episode of BV in the prior | No | х | X | х | х | X | x | x | Х |
| 12 months)? | Yes | х | X | х | х | X | x | x | Х |
| Did the subject have a diagnosis of BV within | No | X | X | X | Х | X | X | X | X |
| the prior 6 months? | Yes | X | X | X | Х | X | X | X | X |
| | Was a new partner | X | X | X | Х | X | X | X | X |
| Subject's most recent sexual partner | Was a male | x | X | X | Х | X | x | X | X |
| Subject's most recent sexual partner | Used a condom | x | X | х | х | X | x | x | Х |
| | N/A | X | X | X | Х | X | X | X | X |
| In the last 30 days, how often did the subject | Always | X | X | X | Х | X | X | X | X |
| use a condom? | Sometimes | X | X | X | X | X | X | X | X |
| | Never | х | X | х | Х | Х | Х | Х | Х |
| In the last 3 months, how often did the subject | Always | x | X | X | X | X | X | X | X |
| use a condom? | Sometimes | X | X | X | X | X | X | X | X |
| | Never | x | X | x | х | x | x | x | Х |

N=Number of subjects in the ITT population who received the specified treatment and has the specified BV status.

Denominator for percentages is the number of subjects in the Amoxicillin group (N) within the specified BV Status category.

Treatment group is the treatment to which the subject was randomized.

Screening Visit 0.

Denominator for percentages is the number of subjects in the Amoxicillin group with male partners in the specified time frame.

Table with similar format:

Table 33: Categorical Baseline Sexual History by Visit 2 BV Status - ITT Population - Placebo Treatment Group

Table 34: Continuous Baseline Sexual History by Visit 2 BV Status - ITT Population – Amoxicillin Treatment Group

| | | Amoxicilli | in (N=X) | | | |
|---|---|---|---|---|---|---|
| Time Frame | Sexual Behavior Characteristic | Statistic | BV by Amsel<br>Criteria<br>(N=X) | BV by Nugent<br>Score<br>(N=X) | BV by Amsel Criteria<br>and Nugent Score<br>(N=X) | No BV by either Amsel<br>or Nugent Score<br>(N=X) |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Days since the subject last had sexual intercourse | Median | x.x | x.x | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of episodes of BV in prior 12 months | Median | x.x | x.x | x.x | x.x |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | Number of times the subject douched or used vaginal preparations or drying agents | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | | Median | x.x | x.x | x.x | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Total number of partners | Median | x.x | x.x | X.X | x.x |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of new partners | Median | x.x | x.x | x.x | x.x |
| In the last 30 | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| days | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of regular partners | Median | x.x | x.x | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| Nu | Number of occasional partners | Median | x.x | x.x | x.x | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of male partners | Median | x.x | x.x | x.x | x.x |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |

Table 34: Continuous Baseline Sexual History by Visit 2 BV Status - ITT Population – Amoxicillin Treatment Group (Continued)

| | | | Amoxicillin (N=X) | | | |
|---|---|---|---|---|---|---|
| Time Frame | Sexual Behavior<br>Characteristic | Statistic | BV by Amsel Criteria<br>(N=X) | BV by Nugent Score<br>(N=X) | BV by Amsel Criteria and<br>Nugent Score<br>(N=X) | No BV by either Amsel<br>or Nugent Score<br>(N=X) |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Total number of partners | Median | X.X | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of new partners | Median | X.X | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| In the last 3 months | Number of regular partners | Median | X.X | X.X | X.X | X.X |
| 1110 110115 | | Minimum, Maximum | x, x | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of occasional partners | Median | X.X | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | X, X | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of male partners | Median | X.X | X.X | X.X | X.X |
| | | Minimum, Maximum | X, X | x, x | x, x | x, x |

N=Number of subjects in the Amoxicillin group with the respective BV Status.

Treatment group is the treatment to which the subject was randomized.

Screening Visit 0.

Table with similar format:

**Table 35:** Continuous Baseline Sexual History by Visit 2 BV Status - ITT Population – Placebo Treatment Group

Table 36: Summary of Categorical Demographic and Baseline Characteristics by Visit 2 BV Status - ITT Population - Amoxicillin Treatment Group

| | | Amo | oxicillin (N=X) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | BV by Amsel Criteria<br>(N=X) | | BV by Nugent Score<br>(N=X) | | BV by Amsel Criteria<br>and Nugent Score<br>(N=X) | | No BV by either Amsel<br>or Nugent Score<br>(N=X) |
| Variable | Characteristic | n | % | n | % | n | % | n | % |
| Sex | Female | х | х | X | x x | х | х | X | х |
| Ethnicity | Not Hispanic or Latino | х | х | X | x | х | х | х | Х |
| | Hispanic or Latino | х | х | X | x | х | х | х | Х |
| | Not Reported | х | х | X | x | х | х | х | Х |
| | Unknown | х | х | X | x | х | х | х | Х |
| Race | American Indian or Alaska Native | х | х | X | x | х | х | х | Х |
| | Asian | х | х | X | x | х | х | х | Х |
| | Native Hawaiian or Other Pacific Islander | х | х | X | x | х | х | х | Х |
| | Black or African American | х | х | X | x | х | х | х | Х |
| | White | х | X | X | x | Х | х | х | Х |
| | Multi-Racial | х | х | х | x | х | х | х | Х |
| | Unknown | х | X | X | x | Х | х | х | Х |

Note: N=Number of Subjects in the ITT population who received Amoxicillin with the respective BV Status at Visit 2.

Treatment group is the treatment to which the subject was randomized.

#### Table with similar format:

Table 37: Summary of Categorical Demographic and Baseline Characteristics by Visit 2 BV Status - ITT Population - Placebo Treatment Group

Table 38: Summary of Continuous Demographic and Baseline Characteristics by Visit 2 BV Status – ITT Population – Amoxicillin Treatment Group

| | Amoxicillin (N=X) | | | | |
|---|---|---|---|---|---|
| Variable | Statistic | BV by Amsel Criteria<br>(N=X) | BV by Nugent Score<br>(N=X) | BV by Amsel Criteria and<br>Nugent Score<br>(N=X) | No BV by either Amsel or<br>Nugent Score<br>(N=X) |
| Age | Mean | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X |
| | Minimum | X | X | X | X |
| | Maximum | X | X | X | X |

Note: N=Number of Subjects in the ITT population who received Amoxicillin with the respective BV Status at Visit 2

Treatment group is the treatment to which the subject was randomized.

#### Table with similar format:

Table 39: Summary of Continuous Demographic and Baseline Characteristics by Visit 2 BV Status – ITT Population – Placebo Treatment Group
Table 40: Summary of Categorical Demographic and Baseline Characteristics by Site - All Enrolled Subjects

| | | at Birr | of Alabama<br>ningham<br>= X) | Wake Forest Health So (N = 2) | iences | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | 0/0 | n | % | n | % |
| Sex | Female | х | XX | X | XX | X | XX |
| Ethnicity | Not Hispanic or Latino | х | xx | X | xx | X | XX |
| | Hispanic or Latino | х | XX | X | xx | X | XX |
| | Not Reported | х | XX | X | xx | X | XX |
| | Unknown | х | XX | X | xx | X | XX |
| Race | American Indian or Alaska Native | х | XX | X | XX | X | XX |
| | Asian | х | XX | X | xx | X | XX |
| | Native Hawaiian or Other Pacific Islander | х | XX | X | xx | X | XX |
| | Black or African American | х | XX | X | xx | X | XX |
| | White | х | XX | X | xx | X | XX |
| | Multi-Racial | х | XX | X | XX | X | XX |
| | Unknown | х | XX | X | xx | X | XX |

N=Number of subjects enrolled at the specified site.

Table 41: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - ITT Population

| | | | xicillin<br>=X) | | cebo<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % |
| Sex | Female | х | xx | х | xx | х | XX |
| Ethnicity | Not Hispanic or Latino | х | xx | х | xx | х | XX |
| | Hispanic or Latino | х | xx | х | xx | х | XX |
| | Not Reported | | xx | х | xx | х | XX |
| | Unknown | х | xx | х | xx | х | XX |
| Race | American Indian or Alaska Native | х | xx | х | xx | х | XX |
| | Asian | х | xx | х | xx | х | XX |
| | Native Hawaiian or Other Pacific Islander | х | xx | х | xx | х | XX |
| | Black or African American | х | xx | х | xx | х | XX |
| | White | х | xx | х | xx | х | XX |
| | Multi-Racial | х | xx | х | xx | X | XX |
| | Unknown | х | xx | х | xx | х | xx |

N=Number of Subjects in the ITT population randomized to the specified treatment group.

Table 42: Summary of Continuous Demographic and Baseline Characteristics by Site—All Enrolled Subjects

| Variable | Statistic | University of Alabama at Birmingham (N = X) | Wake Forest University Health Sciences (N = X) | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Age | Mean | X.X | x.x | x.x |
| | Standard Deviation | X.X | x.x | x.x |
| | Median | X.X | x.x | x.x |
| | Minimum | X | x | x |
| | Maximum | Х | x | x |

Notes: N=Number of subjects enrolled at the specified site.

Table 43: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group - ITT Population

| Variable | Statistic | Statistic Amoxicillin (N=X) | | All Subjects<br>(N=X) |
|---|---|---|---|---|
| Age | Mean | X.X | x.x | X.X |
| | Standard Deviation | X.X | x.x | X.X |
| | Median | X.X | x.x | X.X |
| | Minimum | X | x | X |
| | Maximum | X | x | X |

N=Number of subjects in the ITT population randomized to the specified treatment group.

Table 44: **Categorical Baseline Sexual History by Treatment Group -ITT Population** 

| Sexual Behavior Category | Value | | xicillin<br>=X) | Plac<br>(N= | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % |
| Has the subject ever douched or used vaginal preparations or drying | No | X | X | Х | х | х | Х |
| agents? | Summer's Eve | x | X | Х | Х | х | Х |
| | Rephresh | x | X | Х | Х | х | Х |
| | Vagisil | X | X | Х | х | х | Х |
| | Other | X | X | Х | х | х | Х |
| Does the subjects have a history of recurrent BV (more than one episode of | No | x | X | Х | Х | х | Х |
| BV in the prior 12 months)? | Yes | x | X | Х | Х | х | Х |
| Did the subject have a diagnosis of BV within the prior 6 months? | No | x | X | Х | Х | х | Х |
| Did the subject have a diagnosis of BV within the prior o months: | Yes | X | X | X | X | X | X |
| | Was a new partner | X | X | X | X | X | X |
| Subject's most recent sound mortuon | Was a male | X | X | X | X | X | X |
| Subject's most recent sexual partner | Used a condom | X | X | X | X | X | X |
| | N/A | X | X | х | Х | х | Х |
| In the last 30 days, how often did the subject use a condom? | Always | X | X | х | Х | х | Х |
| | Sometimes | X | X | х | Х | х | Х |
| | Never | х | X | х | х | х | Х |
| In the last 3 months, how often did the subject use a condom? | Always | Х | X | Х | Х | Х | х |
| | Sometimes | Х | X | Х | Х | Х | х |
| | Never | X | X | Х | х | х | Х |

N=Number of Subjects in the ITT population.

Treatment group is the treatment to which the subject was randomized.

Screening Visit 0.

Denominator for percentages is the number of subjects with male partners in the specified time frame.

**Table 45:** Continuous Baseline Sexual History by Treatment Group–ITT Population

| Time Frame | Sexual Behavior<br>Characteristic | Statistic | Amoxicillin<br>(N=X) | Placebo<br>(N=X) | All Subjects (N = X) |
|---|---|---|---|---|---|
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Days since the subject last had sexual intercourse | Median | X.X | X.X | x.x |
| | | Minimum, Maximum | x, x | X, X | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of episodes of BV in prior 12 months | Median | X.X | X.X | x.x |
| | | Minimum, Maximum | x, x | X, X | x, x |
| | Number of times the subject | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | douched or used vaginal | Median | X.X | X.X | x.x |
| | preparations or drying agents | Minimum, Maximum | x, x | X, X | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Total number of partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | X, X | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of new partners | Median | X.X | X.X | x.x |
| the last 30 days | | Minimum, Maximum | x, x | X, X | x, x |
| the last 50 days | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of regular partners | Median | X.X | X.X | x.x |
| | | Minimum, Maximum | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of occasional partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | X, X | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of male partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x |

**Table 45:** Continuous Baseline Sexual History by Treatment Group–ITT Population (Continued)

| Time Frame | Sexual Behavior<br>Characteristic | Statistic | Amoxicillin<br>(N=X) | Placebo<br>(N=X) | All Subjects (N = X) |
|---|---|---|---|---|---|
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Total number of partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of new partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| In the last 3 months | Number of regular partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of occasional partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | x, x | x, x |
| | | Mean (Standard Deviation) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Number of male partners | Median | X.X | X.X | X.X |
| | | Minimum, Maximum | x, x | X, X | x, x |

N=Number of Subjects in the ITT population who randomized to the specified treatment group.

Treatment group is the treatment to which the subject was randomized.

Screening Visit 0.

Table 46: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population – All Sites

| | Amoxicillin<br>(N=X) | | | cebo<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | n | % |
| Any SOC | X | X | X | X | X | X |
| [SOC 1] | X | X | X | X | X | X |
| [SOC 2] | X | X | х | х | Х | х |

N=Number of subjects in the ITT population who received the specified treatment.

Treatment group is the treatment to which the subject was randomized.

n = Number of subjects reporting medical history within the specified SOC.

A subject is only counted once per SOC.

#### Tables with Similar Format:

Table 47: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population – University of Alabama at Birmingham

Table 48: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group - ITT Population – Wake Forest University Health Sciences

Table 49: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - All Subjects

| | | All Subjec | ts (N=X) | | | | |
|---|---|---|---|---|---|---|---|
| WHO Drug Code | WHO Drug Code | | oxicillin<br>N=X) | | cebo<br>=X) | All Subjects (N=X) | |
| Level 1, Anatomic Group | Level 2, Therapeutic Subgroup | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | x | X | X | X | X | X |
| [ATC Level 1 - 1] | Any | x | X | х | X | Х | X |
| | [ATC 2 - 1] | x | X | x | X | X | X |
| | [ATC 2 - 2] | x | X | x | X | X | X |
| | [ATC 2 - 3] | x | x | x | x | x | X |
| [ATC Level 1 – 2] | Any | x | X | X | X | X | X |
| | [ATC 2 - 1] | x | X | X | x | X | X |
| | [ATC 2 - 2] | X | X | X | x | X | X |
| N. N. J. C. Li. et al. G.C. | [ATC 2 - 3] | X | X | X | X | X | X |

N= Number of subjects in the Safety population who received the specified treatment.

#### Tables with Similar Format:

Table 50: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - University of Alabama at Birmingham

Table 51: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group - Safety Population - Wake Forest University Health Sciences

n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

Table 52: Proportion of Subjects Reporting Treatment Related Adverse Events Following the First Dose of Treatment through Visit 2 by Treatment Group – Safety Population

| Treatment<br>Group | Number of<br>Subjects with AEs<br>n | Number of<br>Subjects<br>N | Proportion of<br>Subjects with AEs | Proportion of<br>Subjects with AEs<br>95% CI | Difference in Proportion of<br>Subjects with AEs between<br>Amoxicillin and Placebo | Difference in Proportion of Subjects with<br>AEs between Amoxicillin and Placebo<br>95% CI | P-value |
|---|---|---|---|---|---|---|---|
| Amoxicillin | Х | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Placebo | Х | X | 0.xx | 0.xx, 0.xx | | | |
| All Subjects | Х | X | 0.xx | 0.xx, 0.xx | | | |

The denominator for proportions is based on the number of subjects who received the specified treatment. 95% CI = 95% Blaker confidence interval.

P-value from the Fisher's exact two-sided test at the .05 level of significance.

Table 53: Proportion of Subjects Discontinuing Treatment Early Due to Adverse Events by Treatment Group – Safety Population

| Treatment<br>Group | Number of<br>Subjects with AEs<br>n | Number of<br>Subjects<br>N | Proportion of Subjects Discontinuing Early due to AEs | Proportion of Subjects Discontinuing Early due to AEs 95% CI | Difference in Proportion of<br>Subjects Discontinuing Early due<br>to AEs between Amoxicillin and<br>Placebo | Difference in Proportion of Subjects Discontinuing Early due to AEs between Amoxicillin and Placebo 95% CI | P-value |
|---|---|---|---|---|---|---|---|
| Amoxicillin | X | X | 0.xx | 0.xx, 0.xx | 0.xx | 0.xx, 0.xx | 0.xxx |
| Placebo | X | X | 0.xx | 0.xx, 0.xx | | | |
| All Subjects | x | X | 0.xx | 0.xx, 0.xx | | | |

The denominator for proportions is based on the number of subjects who received the specified treatment.

<sup>95%</sup> CI = 95% Blaker confidence interval.

P-value from the Fisher's exact two-sided test at the .05 level of significance.

Table 54: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population

| MedDRA System Organ | MedDRA Preferred | Amoxicillin<br>(N=X) | | | Placebo<br>(N=X) | | | | All Subjects<br>(N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class | Term | n | % | 95% CI | Events | n | % | 95% CI | Events | n | % | 95% CI | Events |
| Any SOC | Any PT | X | х | x, x | X | X | х | x, x | X | X | х | x, x | X |
| [SOC 1] | Any PT | Х | х | x, x | X | х | х | x, x | X | х | х | x, x | X |
| | [PT 1] | Х | х | x, x | X | х | х | x, x | X | х | х | x, x | Х |
| | [PT 2] | Х | х | x, x | X | х | х | x, x | X | х | х | x, x | X |
| [SOC 2] | Any PT | X | х | x, x | X | X | х | x, x | x | х | х | x, x | X |
| | [PT 1] | X | х | x, x | X | X | х | x, x | x | х | х | x, x | X |
| | [PT 2] | Х | х | x, x | х | х | х | x, x | x | х | х | x, x | x |

N = Number of subjects in the Safety Analysis Population who received the specified treatment.

<sup>95%</sup> CI = 95% Blaker confidence interval.

This table presents number and percentage of subjects.

A subject is only counted once per PT/timepoint.

Table 55: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity and Relationship - Safety Population

| | | | All Subjects (N = X) | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Rel | ated | Not R | Related | Total | |
| | | | n | % | n | % | n | % |
| Any SOC | Any PT | Any Severity | Х | Х | Х | Х | Х | Х |
| | | Mild | Х | Х | Х | Х | Х | X |
| | | Moderate | Х | Х | Х | Х | Х | X |
| | | Severe | х | х | х | х | х | X |
| [SOC 1] | Any PT | Any Severity | Х | Х | Х | Х | X | X |
| | | Mild | Х | Х | Х | Х | X | X |
| | | Moderate | х | х | х | х | х | X |
| | | Severe | х | х | х | х | х | X |
| | [PT 1] | Any Severity | х | х | х | х | х | X |
| | | Mild | х | Х | Х | х | X | X |
| | | Moderate | х | Х | X | X | X | X |
| | | Severe | х | х | х | X | x | X |

N = Number of subjects in the Safety Analysis Population

This table presents number and percentage of subjects as well as number of events.

For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

Table 56: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - Safety Population

| | | | | Amoxicillin<br>(N = X) | | | | | Placebo<br>(N = X) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Rel | ated | Not R | Not Related | | Total | | Related | | Not Related | | Total |
| | | | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | Any Severity | x | х | х | х | х | х | х | х | х | х | х | х |
| | | Mild | x | х | х | х | х | х | х | х | х | х | х | х |
| | | Moderate | x | X | х | х | х | х | х | х | х | х | х | x |
| | | Severe | x | х | х | х | х | х | x | х | х | х | х | x |
| [SOC 1] | Any PT | Any Severity | x | х | х | х | х | х | х | х | х | х | х | х |
| | | Mild | X | х | х | х | х | х | х | х | х | х | х | х |
| | | Moderate | X | х | х | х | х | х | х | х | х | х | х | х |
| | | Severe | X | х | х | х | х | х | х | х | х | х | х | х |
| | [PT 1] | Any Severity | X | х | х | х | х | х | х | х | х | х | х | х |
| | | Mild | X | х | х | х | х | х | х | х | х | х | х | х |
| | | Moderate | X | х | х | х | х | х | х | х | х | х | х | х |
| | ubjects in the Safety A | Severe | X | Х | Х | Х | Х | Х | х | х | Х | Х | Х | Х |

N = Number of subjects in the Safety Analysis Population who received the specified treatment.

This table presents number and percentage of subjects as well as number of events.

For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

Table 57: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class, Preferred Term, and Treatment Group - Safety Population

| Preferred Term | MedDRA System Organ Class | Amoxicillin<br>(N=X) | | | Placebo<br>(N=X) | | | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Events | | | | | | | | | | |
| All | All | x | x | x | x | х | x | X | x | X |
| PT1 | SOC1 | x | х | x | х | х | X | X | x | X |
| Etc. | Etc. | x | х | x | х | х | X | X | x | X |
| Non-serious Adverse Events | | | | | | | | | | |
| All | All | x | x | x | x | х | x | X | x | X |
| PT1 | SOC1 | x | х | x | х | х | x | x | x | х |
| Etc | Etc | X | х | X | х | х | X | X | Х | X |

N = number of subjects in the Safety Population who received the specified treatment.

n= number of subjects reporting event.

This table presents number and percentage of subjects as well as number of events.

### Table 58: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | Study<br>Day | Severity | Relationship to<br>Study Treatment | In Not Related,<br>Alternative Etiology | Action Taken with Study Treatment | Subject Discontinued<br>Due to AE | Outcome | MedDRA System<br>Organ Class | MedDRA<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Treatment Group: , AE Number: | | | | | | | | | |
| xxxxxxx | xx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments:x | xxxxxxxx | ίχ | | | | | | | |
| Subject ID:, | Subject ID: , Treatment Group: , AE Number: | | | | | | | | |
| xxxxxxx | xx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments:x | XXXXXXXXX | ΚX | | | | | | | |

### **Table 59:** Listing of Serious Adverse Events

| Adverse<br>Event | Study Day the<br>Event Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship to Study<br>Treatment | In Not Related,<br>Alternative Etiology | Action Taken with<br>Study Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Treatment Group: , AE Number: | | | | | | | | | | |
| xxxxxx | xx | xxxxxx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments: x | Comments: xxxxxxxxxxx | | | | | | | | | |
| Subject ID: | , Treatment Grou | p: , AE Numb | er: | | | | | | | |
| xxxxxx | xx | xxxxx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | XXXXX |
| Comments: x | Comments: xxxxxxxxxxx | | | | | | | | | |

# APPENDIX 2. FIGURE MOCK-UPS

## LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 84 |
|---|---|---|
| Figure 2: | Nugent Scores by Visit and Treatment Group - ITT Population | 85 |
| Figure 3: | Nugent Scores by Visit and Treatment Group - PP Population | 85 |
| Figure 4: | Frequency of Adverse Events by MedDRA System Organ Class and Severity | 86 |
| Figure 5: | Incidence of Adverse Events by MedDRA System Organ Class and Maximum Severity | 87 |

Figure 1: CONSORT Flow Diagram





Figure 2: Nugent Scores by Visit and Treatment Group - ITT Population

Figures with similar format:

Figure 3: Nugent Scores by Visit and Treatment Group - PP Population



Figure 4: Frequency of Adverse Events by MedDRA System Organ Class and Severity

Group A will be Amoxicillin and Group B will be Placebo.

Figure 5: Incidence of Adverse Events by MedDRA System Organ Class and Maximum Severity



Group A will be Amoxicillin and Group B will be Placebo.

# APPENDIX 3. LISTINGS MOCK-UPS

## **LISTINGS**

| Listing 1: | Subjects Excluded from Analysis Populations | 91 |
|---|---|---|
| Listing 2: | Subjects Whose Assigned Treatment Group Does Not Match Their Randomized Treatment Group | 92 |
| Listing 3: | Early Terminations or Discontinued Subjects-All Enrolled Subjects | 93 |
| Listing 4: | Subject-Specific Protocol Deviations-All Enrolled Subjects | 94 |
| Listing 5: | Non-Subject-Specific Protocol Deviations | 95 |
| Listing 6: | Individual Efficacy Response Data- All Enrolled Subjects | 96 |
| Listing 7: | Individual Clinical Laboratory Results- GV Negative Subjects at Screening | 97 |
| Listing 8: | Demographic Data - All Enrolled Subjects | 98 |
| Listing 9: | Demographic Data - GV Negative Subjects | 98 |
| Listing 10: | Sexual History at Screening - All Enrolled Subjects | 99 |
| Listing 11: | Sexual History at Screening - GV Negative Subjects | 99 |
| Listing 12: | Sexual Behavior History at Screening - All Enrolled Subjects | 100 |
| Listing 13: | Sexual Behavior History at Screening – GV Negative Subjects | 100 |
| Listing 14: | Sexual Behavior History at Screening - Last 3 Months - All Screened Subjects | 101 |
| Listing 15: | Sexual Behavior History at Screening - Last 3 Months – GV Negative Subjects | 101 |
| Listing 16: | Interim Sexual Behavior History - All Enrolled Subjects | 102 |
| Listing 17: | Pre-Existing Medical Conditions - All Enrolled Subjects | 103 |
| Listing 18: | Concomitant Medications - All Enrolled Subjects | 104 |
| Listing 19: | Birth Control Methods - All Enrolled Subjects | 105 |
| Listing 20: | Unsolicited Adverse Events - Safety Population | 106 |
| Listing 21: | Pregnancy Reports – Maternal Information | 107 |
| Listing 22: | Pregnancy Reports – Gravida and Para | 108 |
| Listing 23: | Pregnancy Reports – Live Birth Outcomes | 109 |
| Listing 24: | Pregnancy Reports – Still Birth Outcomes | 110 |
| Listing 25: | Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 111 |
| Listing 26: | Pelvic Exam Findings - All Enrolled Subjects | 112 |

| Statistical Analysis Plan - DMID Protocol: 16-0073 | Version 1.0 |
|-------------------------------------------------------------|-------------|
| | 27FEB2019 |
| Listing 27: KOH Saline Microscopy - All Enrolled Subjects | 113 |
| Listing 28: BV Microbiology Results - All Screened Subjects | 114 |

## **Listing of Subjects Receiving Investigational Product**

(not included in SAP, but this is a placeholder for the CSR)

**Listing 1:** Subjects Excluded from Analysis Populations

| Actual Treatment<br>Group | Randomized<br>Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason(s) Subject Excluded |
|---|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Visit x] | Yes/No | xxxxx |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Visit x] | Yes/No | xxxxx |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Visit x] | Yes/No | xxxxx |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. If "Yes" the population in which data were removed will be listed in parenthesis. "No" indicates that no data were available for inclusion in the analysis.

- 1. Sort order will be actual treatment group, Subject ID
- 2. Reasons Subject Excluded should match the same verbiage that is used on the Analysis population tables
- 3. If all subjects received the correct treatment, only display "Treatment Group".

### Listing 2: Subjects Whose Assigned Treatment Group Does Not Match Their Randomized Treatment Group

| Subject ID | Treatment Group at Randomization | Treatment Actually Received |
|---|---|---|
| xxxxxx | Amoxicillin/Placebo | Amoxicillin/Placebo |
| xxxxxx | Amoxicillin/Placebo | Amoxicillin/Placebo |

Implementation Note:

1. Sort order is Subject ID.

**Listing 3:** Early Terminations or Discontinued Subjects-All Enrolled Subjects

| Actual Treatment Group | Randomized<br>Treatment Group | Subject ID | Category | Study Day Corresponding to Early<br>Termination/Treatment<br>Discontinuation/Completion | Reason for Early Termination/<br>Treatment Discontinuation |
|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo xxxxxxx Early Termination/Treatment Discontinuation/Completion | | xx | xxxxxxxxxxxxx | |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxxx | Early Termination/Treatment<br>Discontinuation/Completion | xx | |

- 1. Sort order will be by Actual Treatment Group, Subject ID, Category
- 2. If all subjects received the correct treatment, only display "Treatment Group".
- 3. Category will be "Early Termination", "Completion" or "Treatment Discontinuation". If a subject discontinued treatment, they will have two records.
- 4. In the "Reason" column, concatenate any "specify" fields, including AE number and DV number.

**Listing 4:** Subject-Specific Protocol Deviations-All Enrolled Subjects

| Deviation<br>Number | Study<br>Day | Deviation<br>Description | Deviation Category | Reason for<br>Deviation | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resulted in<br>AE? | Deviation Resulted<br>in Subject<br>Termination? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|
| Actual Treatme | Actual Treatment Group: , Randomized Treatment Group: , Subject ID: | | | | | | | | |
| xx | xx | xxxxxxx | xxxxxxxxxx | xxxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | xxxxxxxxxx |
| xx | xx | xxxxxxx | xxxxxxxxxx | xxxxxxx | Yes/No | Yes/No | Yes/No | Yes/No | |

Note: Deviation description column will contain all subfields concatenated together

- 1. Sort order will be by Actual Treatment Group, Subject ID, Deviation Number
- 2. In the Deviation Category column concatenate any specify fields
- 3. In the Reason for Deviation column concatenate any specify fields.

**Listing 5:** Non-Subject-Specific Protocol Deviations

| Site | Deviation | Start Day | End Day | Reason for<br>Deviation | Deviation Resulted<br>in Subject<br>Termination? | Deviation Affected<br>Product Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | XX | XX | XXXX | Yes/No | Yes/No/NA | XXXX | XXXX | XXXX |
| XXXX | xxxx | XX | XX | XXXX | Yes/No | Yes/No/NA | XXXX | xxxx | Xxxx |

Note: Deviation description column will contain all subfields concatenated together

- 1. Sort order will be by Site Name, Start Date
- 2. In the Deviation Category column concatenate any specify fields
- 3. In the Reason for Deviation column concatenate any specify fields.

### **Listing 6:** Individual Efficacy Response Data- All Enrolled Subjects

| Study<br>Day | Trichomonas<br>NAAT Result | Vaginal pH | Amine ("whiff") test on<br>KOH wet mount | Clue Cells | Amsel Criteria | Amsel Criteria Nugent Score | | <b>GV Eradication Status</b> |
|---|---|---|---|---|---|---|---|---|
| Actual Treatment Group: , Randomized Treatment Group: Subject ID: | | | | | | | | |
| x | Negative/Positive | xx.x | Negative/Positive | Negative/ <20%/<br>>=20% | х | х | Xx10 <sup>x</sup> /Negative/<br>LLOQ/ULOQ | Eradicated/Not<br>Eradicated/Not<br>Evaluable |

- 1. Sort order is actual treatment group, Subject ID, Study Day.
- 2. If all subjects received the correct treatment, only display "Treatment Group".
- 3. Trichomonas NAAT only performed at screening visit, populate cells at later visits with "—"
- 4. GV Eradication Status is only available for Visit 2, display "—" for Visit 1.

### Listing 7: Individual Clinical Laboratory Results- GV Negative Subjects at Screening

| Site | Subject ID | Trichomonas NAAT<br>Result | Vaginal pH | Amine ("whiff") test on<br>KOH wet mount | Clue Cells | Amsel Criteria | Nugent Score | GV NAAT Result |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxx | Negative/Positive | XX.X | Negative/Positive | xx | x | X | Xx10 <sup>x</sup> /Negative/<br>LLOQ/ULOQ |

Implementation Notes:

1. Sort order is Subject ID.

**Listing 8:** Demographic Data - All Enrolled Subjects

| Screen Failure? | Actual Treatment Group | Randomized Treatment Group | Subject ID | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|---|
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | XXXXXX | XX | xxxxxx | xxxxxx |
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | xxxxxx | xxxxxx |
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | xxxxxx | xxxxxx |

- 1. Sort order will be by screen failure, Actual Treatment Group, Subject ID
- 2. For the Race column, if a subject is Multi-Racial, all races will be listed, separated by a comma
- 3. If subject was a screen failure, populate actual treatment group and randomized treatment group with "—"
- 4. If all subjects received the correct treatment, only display "Treatment Group".

### Listing with similar format:

### **Listing 9:** Demographic Data - GV Negative Subjects

**Listing 10:** Sexual History at Screening - All Enrolled Subjects

| Screen<br>Failure? | Actual Treatment<br>Group | Randomized<br>Treatment Group | Subject<br>ID | Day of Subjects<br>Last Menstrual<br>Period | Ever Douched or Used<br>Vaginal Preparations or<br>Drying Agents? | If Yes, Specify Product | Number of Times Douched or Used<br>Vaginal Preparations or Drying<br>Agents in the last 30 Days |
|---|---|---|---|---|---|---|---|
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | Yes/No | Summer's<br>Eve/Rephresh/Vagisil/Other(specify) | xx |
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | xx | Yes/No | Summer's<br>Eve/Rephresh/Vagisil/Other(specify) | xx |

- 1. Sort order will be by screen failure, Actual Treatment Group, Subject ID
- 2. If the subject has used "other" Vaginal Preparations or Drying Agents, list the specify field in the cell
- 3. If subject was a screen failure, populate actual treatment group and randomized treatment group with "—"
- 4. If all subjects received the correct treatment, only display "Treatment Group".

#### Listing with similar format:

### **Listing 11:** Sexual History at Screening - GV Negative Subjects

**Listing 12:** Sexual Behavior History at Screening - All Enrolled Subjects

| | | | | | | | | Most Recent Sexual<br>Partner | | | In the Last 30 Days | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Screen<br>Failure? | Actual<br>Treatment<br>Group | Randomized<br>Treatment<br>Group | Subject<br>ID | | of<br>episodes<br>of BV in | Had a diagnosis of BV within the prior 6 months | Day Since<br>the Subject<br>Last had<br>Vaginal<br>Sexual<br>Intercourse | A New<br>Partner? | A<br>Male? | Was a condom used? | Total<br>Number<br>of<br>Sexual<br>Partners | Number<br>of New<br>Partners | Number<br>of<br>Regular<br>Partners | Number of<br>Occasional<br>Partners | Number<br>of Male<br>Partners | How Often<br>was a<br>condom<br>used? |
| Y/N | Amoxicillin/<br>Placebo | Amoxicillin/<br>Placebo | xxxxxx | Yes/No | xx | Yes/No | XX | Yes/No | Yes/No | Yes/No | xx | xx | xx | xx | XX | Always/<br>Sometimes/<br>Never |
| Y/N | Amoxicillin/<br>Placebo | Amoxicillin<br>/Placebo | xxxxxx | Yes/No | xx | Yes/No | XX | Yes/No | Yes/No | Yes/No | xx | xx | xx | xx | XX | Always/<br>Sometimes/<br>Never |

- 1. Sort order will be by Screen failure, Actual Treatment Group, Subject ID
- 2. If subject was a screen failure, populate actual treatment group and randomized treatment group with "—"
- 3. If all subjects received the correct treatment, only display "Treatment Group".

### Listing with similar format:

## **Listing 13:** Sexual Behavior History at Screening – GV Negative Subjects

Listing 14: Sexual Behavior History at Screening - Last 3 Months - All Screened Subjects

| | | | | | In the Last 3 Months | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Screen<br>Failure? | Actual Treatment<br>Group | Randomized Treatment<br>Group | Subject<br>ID | Total Number of<br>Sexual Partners | Number of<br>New Partners | Number of<br>Regular Partners | - ( | | How Often was a condom used? |
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | xx | XX | XX | XX | XX | Always/Sometimes/Never |
| Y/N | Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | xx | XX | XX | XX | XX | Always/Sometimes/Never |

- 1. Sort order will be by Screen Failure, Actual Treatment Group, Subject ID
- 2. If subject was a screen failure, populate actual treatment group and randomized treatment group with "—"
- 3. If all subjects received the correct treatment, only display "Treatment Group".

### Listing with similar format:

### Listing 15: Sexual Behavior History at Screening - Last 3 Months - GV Negative Subjects
**Listing 16:** Interim Sexual Behavior History - All Enrolled Subjects

| | | | | Since Last Visit | | | | |
|---|---|---|---|---|---|---|---|---|
| Actual Treatment<br>Group | Randomized Treatment<br>Group | Subject<br>ID | Study Day | Total Number of<br>Sexual Partners | Number of New<br>Partners | Number of Regular<br>Partners | Number of Occasional<br>Partners | Number of Male<br>Partners |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | XX | XX | XX | xx | XX |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | XX | XX | XX | xx | XX |

- 1. Sort order will be by Actual Treatment Group, Subject ID
- 2. If all subjects received the correct treatment, only display "Treatment Group".

## **Listing 17: Pre-Existing Medical Conditions - All Enrolled Subjects**

| Actual Treatment Group | Randomized Treatment Group | Subject ID | MH Number | Medical History<br>Term | Condition<br>Start Day | Condition End<br>Day | MedDRA System<br>Organ Class | MedDRA<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XXX | xxxxxx | XX | xx | xxxxxx | xxxxxx |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XXX | xxxxxx | XX | xx | xxxxxx | xxxxxx |

- 1. Sort order is Actual Treatment Group, Subject ID, MH Number.
- 2. "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). Rather than use exact study days, categorize as follows:
  - > 5 years prior to enrollment
  - 1-5 years prior to enrollment
  - -1-12 months prior to enrollment
  - -Within 1 month of enrollment
  - -During Study
  - -If Ongoing at the end of the study, display "Ongoing' in the "Condition End Day" column.
  - -If ending is unknown at the end of the study, display "Unknown" in the "Condition End Day" column.
- 3. If all subjects received the correct treatment, only display "Treatment Group".

**Listing 18:** Concomitant Medications - All Enrolled Subjects

| Actual Treatment<br>Group | Randomized<br>Treatment Group | Subject ID | Concomitant<br>Medication<br>Number | Medication | Medication<br>Start Day | Medication<br>End Day | Indication | Taken for an AE?<br>(AE Description; AE<br>Number) | Taken for a condition on Medical<br>History?<br>(MH Description; MH Number) |
|---|---|---|---|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | xxxxxx | XX | XX | xxxxxx | Yes/No<br>xxxxx; xx | Yes/No<br>xxxxx; xx |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | XX | xxxxxx | XX | XX | xxxxxx | Yes/No<br>xxxxx; xx | Yes/No<br>xxxxx; xx |

- 1. Sort order is actual treatment group, Subject ID, concomitant medication number.
- 2. 'Medication Start Day' and 'Medication End Day' are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact days, categorize as follows:
  - > 5 years prior to enrollment
  - 1- 5 years prior to enrollment
  - 1-12 months prior to enrollment.
  - For 'Medication End Day', if medication is Ongoing, display 'Ongoing' in the Medication End Day' column.
  - For 'Medication End Day', if end of medication is unknown, display 'Unknown' in the 'Medication End Day' column.
- 3. If a Medication is taken for an AE, then concatenate the conmed with the Advere Events by AENUM and report the AETERM, plus the AE Number.
- 4. If a Medication is taken for an MH, then concatenate the conmed with the Medical History event by MHNUM and report the MHTERM, plus the MH Number.
- 5. Include the birth control information in this dataset. The birth control information is coming from the RP/SUPPRP or BC1 dataset.
- 6. If all subjects received the correct treatment, only display "Treatment Group".

## **Listing 19:** Birth Control Methods - All Enrolled Subjects

| Actual Treatment Group | Randomized Treatment Group | Subject ID | Is the subject of childbearing potential? | Method of Birth Control | Start Day | End Day |
|---|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | Yes/No | xxxxxx | XX | XX |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | Yes/No | xxxxxx | XX | xx |

- 1. Sort order is actual treatment group, Subject ID.
- 2. If all subjects received the correct treatment, only display "Treatment Group".
- 3. Subject may have multiple records of Method of Birth Control.

## **Listing 20:** Unsolicited Adverse Events - Safety Population

| Adverse<br>Event | Study<br>Day | Severity | SAE? | Relationship to<br>Study Treatment | In Not Related,<br>Alternative Etiology | Action Taken with<br>Study Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Actual Treat | ment Grou | p: , Random | ized Treatr | nent Group: , Subject I | D: , AE Number: | | | | | |
| xxxxxx | xx | xxxxxx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments: x | xxxxxxxxx | XX | | | | | | | | |
| Actual Treat | ment Grou | p: , Random | ized Treatr | nent Group: , Subject I | D: , AE Number: | | | | | |
| xxxxxx | xx | xxxxxx | xxxxxx | xxxxxx | xxxxx | xxxxxx | Y/N | xxxxx | xxxxx | xxxxx |
| Comments: x | xxxxxxxxx | xx | | | | | | | | |

Note: For additional details about SAEs, see Table X.

- 1. Sort order is actual treatment group, Subject ID, AE Number.
- 2. If all subjects received the correct treatment, only display "Treatment Group".

**Listing 21:** Pregnancy Reports – Maternal Information

| Actual<br>Treatment<br>Group | Actual<br>Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal Complications During Labor, Delivery, or Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Amoxicillin<br>/Placebo | Amoxicillin<br>/Placebo | xxxxxxxx | xx | xx | xxx | xxx | xxx | xxx | Y/N | Y/N | Y/N | Y Y/N /N |
| Amoxicillin<br>/Placebo | Amoxicillin<br>/Placebo | xxxxxxxx | XX | XX | xxx | xxx | xxx | xxx | Y/N | Y/N | Y/N | Y Y/N /N |

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

- 1. Sort order is actual treatment group, Subject ID
- 2. If all subjects received the correct treatment, only display "Treatment Group".

**Listing 22:** Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>Preterm<br>Births | Very<br>Preterm<br>Births | Early<br>Preterm<br>Births | Late<br>Preterm<br>Births | Early<br>Term<br>Births | Full<br>Term<br>Births | Late<br>Term<br>Births | Post<br>Term<br>Births | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly with<br>Previous<br>Pregnancy? |
| xxxxxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | Y/N |
| xxxxxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | Y/N |

Note: Gravida includes the current pregnancy, para events do not.

**Listing 23:** Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress<br>During<br>Labor and<br>Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXX | xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | Y/N | XXX |
| xxxxxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | Y/N | xxx |

Note: Congenital Anomalies are included in the Adverse Event listing.

# **Listing 24:** Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome (for<br>this Fetus) | Fetal Distress<br>During Labor<br>and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord<br>pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for<br>Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XX | XXX | xxxxxxx | Y/N | xxxxxxx | xxx | XXX | XX | Y/N | Y/N | xxxxxxx |

# **Listing 25:** Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|
| xxxxxx | xx | xxx | xxxxx | XXXX | Y/N | xxxxxxx |

### **Listing 26:** Pelvic Exam Findings - All Enrolled Subjects

| Actual Treatment<br>Group | Randomized Treatment<br>Group | Subject ID | Study Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; AE Number) |
|---|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxxx | xxx | xxxxxxxx | xxxxxxxx | Yes/No<br>xxxxxx; xx |

- 1. Sort order is actual treatment group, Subject ID, Study Day.
- 2. If all subjects received the correct treatment, only display "Treatment Group".
- 3. Only abnormal findings will be presented.
- 4. If the physical exam was reported as an AE, then concatenate the Physical exam with the Adverse Events by AENUM and report the AETERM, plus the AE Number

**Listing 27:** KOH Saline Microscopy - All Enrolled Subjects

| Actual Treatment<br>Group | Randomized Treatment<br>Group | Subject<br>ID | Yeast Forms Identified (buds or hyphal elements)? | Quantity of Yeast forms identified? | Wet mount slide for the microscopic observation of <i>T. vaginalis</i> obtained? | T. vaginalis Present? |
|---|---|---|---|---|---|---|
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | Y/N | Rare (<5/HPF)/<br>Few (5-10 HPF)/<br>Numerous (>10HPF) | Y/N | Absent/Present |
| Amoxicillin/Placebo | Amoxicillin/Placebo | xxxxxx | Y/N | Rare (<5/HPF)/<br>Few (5-10 HPF)/<br>Numerous (>10HPF) | Y/N | Absent/Present |

- 1. Sort order is Actual Treatment Group, Subject ID
- 2. If all subjects received the correct treatment, only display "Treatment Group".

## **Listing 28:** BV Microbiology Results - All Screened Subjects

| Screen<br>Failure | Subject ID | Randomized Treatment<br>Group | Actual Treatment Group | Visit | Study<br>Day | Nugent Lactobacillus<br>spp. Score | Nugent Gardnerella/Bateriodes<br>Score | Mobiluncus<br>Score |
|---|---|---|---|---|---|---|---|---|
| Y/N | xxxxxx | Amoxicillin/Placebo | Amoxicillin/Placebo | 00 | XX | xxxxxxxx | XXXXXXXX | xxxxxxxx |
| | | | | 02 | XX | xxxxxxxx | XXXXXXXX | xxxxxxxx |

- 1. Sort order is Screen Failure, Actual Treatment Group, Subject ID, Study Day.
- 2. Unscheduled visits will be included
- 3. If subject was a screen failure, populate actual treatment group and randomized treatment group with "—"
- 4. If all subjects received the correct treatment, only display "Treatment Group".